



STATISTICAL ANALYSIS PLAN Protocol: RB244-001


# STATISTICAL ANALYSIS PLAN PHASE II

**VERSION: 1.0** 

**DATE:** 

**February 14, 2019** 

## **BASED ON:**

Protocol Version 4.0 Date:07-Jan-19

Data Management Plan Final Version 1.0 Date: 12-Apr-18

# **Study Drug:**

**B244** Topical Application

# **Protocol Number:**

RB244-001

# **Study Title:**

Vehicle-Controlled, Double-Blind, Randomized Phase II Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects with Mild to Moderate Rosacea.

# **Sponsor:**

AOBiome, LLC

125 Cambridgepark Drive

Cambridge, MA 02140

NCT03590366







Protocol: RB244-001

STATISTICAL ANALYSIS PLAN

Version 1 14-Feb-19


# STATISTICAL ANALYSIS PLAN REVIEW AND APPROVAL

| This Statistical Analysis Plan has been prepared in accordance with team reviewers' specifications. | |
|---|---|
| Prepared by: Rahul-Paul Choudhury, Lead Bio-Statistician | 19 FEB 2019<br>Date |
| Statistical Review: Jose Nabut, Sr. Specialist Bio-Statistician | 19Feb 2019<br>Date |
| Sponsor Review: | |
| Judith Ng-Cashin, M.D. Chief Medical Officer | 14 Feb 2019<br>Date |
| Spiros Jamas, Sc. D., SVP of Therapeutic Development | Feb 14th 2019 Date |





Version 1

14-Feb-19

Protocol: RB244-001 STATISTICAL ANALYSIS PLAN

# **PROTOCOL SYNOPSIS**

| Study Title | A Vehicle-Controlled, Double-Blind, Randomized Phase II Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects with Mild to Moderate Rosacea. |
|---|---|
| Protocol Number | RB244-001 |
| <b>Development Phase</b> | Phase II |
| Type of Study | Safety Analysis and Superiority of the Study drug over Vehicle |
| Study Medications | <ol> <li>B244 Topical Spray (Test formulation), manufactured by<br/>AOBiome Therapeutics.</li> <li>Vehicle of test product manufactured by AOBiome<br/>Therapeutics.</li> </ol> |
| Name of Active<br>Ingredient | B244 |
| Route of administration | Topical application |
| Sponsor | AOBiome, LLC,125 Cambridgepark Drive, |
| | Cambridge, MA 02140 |
| Study Objectives | PRIMARY |
| | To assess the safety and tolerability of B244 applied twice daily (BID) to the face for 8 weeks in subjects with mild to moderate rosacea. |
| | EXPLORATORY |
| | To assess the efficacy of B244 in subjects with mild to moderate rosacea. |
| | <ul> <li>Proportion of subjects with IGA improvement at Week 8 relative to baseline</li> <li>Proportion of subjects with CEA improvement at Week 8 relative to baseline</li> <li>Change in IGA from Baseline to Week 8</li> <li>Change in CEA from Baseline to Week 8</li> <li>Proportion of Subjects with improvement in IGA or</li> </ul> |



Protocol: RB244-001

CLINICAL RESEARCH OPTIMIZED™



Version 1

| Protocol: RB244-001 | STATISTICAL ANALYSIS PLAN | version i |
|---|---|---|
| | <ul> <li>CEA at Week 1, Week 4, and Week 12.</li> <li>Change in Skindex 16 patient reported outcome from Baseline to Week 1, Week 4, Week 8, and Week 12.</li> <li>Proportion of subjects with change in PSA at Week 1, Week 4, Week 8 and Week 12 from Baseline.</li> <li>Evaluation of Telangiectasia Score at Baseline/Day1 and Week 8</li> </ul> | |
| Study Design | This is a Prospective, Vehicle Controlled, Double Blind, Mult Randomized Phase II trial, comparing the effect of twice dail application for 8 weeks vs. vehicle application on treatment of moderate rosacea. • We will enroll approximately 130 subjects and complete | y B244<br>mild to |
| | <ul> <li>we will cliffly approximately 130 subjects and complete subjects.</li> <li>At Screening and Baseline: <ul> <li>All subjects must have diagnosis of mild to mode Rosacea.</li> <li>Subjects must have IGA score of 2-3 and CEA so</li> </ul> </li> </ul> | erate |
| | <ul> <li>2-3 to qualify for the study.</li> <li>After screening and recruitment, participants will be randomized to active or vehicle application for 8 weeks.</li> <li>Subjects will apply a total of 4 pumps of IP per application the face twice-a-day</li> </ul> | |
| | <ul> <li>Randomization will be 1:1 B244 to Vehicle.</li> <li>Subjects will be provided with cleanser and moisturizer to for the duration of the study</li> <li>All B244 randomized subjects will be treated at the dose 4x109 cells/ml via spray application</li> </ul> | |
| | <ul> <li>Screening period will occur at Days -21 to -1</li> <li>Washout will occur after Screening visit (Days - 14 to -1</li> <li>Randomization will occur during the baseline visit for th Efficacy will be assessed using Investigator Global Asse (IGA) score, Clinician's Erythema Assessment (CEA) screening visit (Days - 14 to -1</li> <li>Randomization will occur during the baseline visit for the Efficacy will be assessed using Investigator Global Asse (IGA) score, Clinician's Erythema Assessment (CEA) score and patient reported Skindex 16.</li> </ul> | e study<br>ssment<br>core, |
| | <ul> <li>Clinical assessments of response to treatment will be ma Week 1(Day 7), Week 4 (Day 28), and Week 8 (Day 56)</li> <li>At Baseline visit, subjects will receive a kit containing the product. Each bottle will be used for 2 weeks. At Week subjects will return the used bottles from the kit and will issued a new kit of drug product to be used from Week 4 through Week 8.</li> </ul> | ne drug<br>4,<br>be |
| | Subjects will stop applying investigational product at We and will return investigational product at that visit. | eek 8 |

STATISTICAL ANALYSIS PLAN



Protocol: RB244-001





Version 1

| ~ ~ | STATISTICAL ANALYSIS PLAN VERSION 1 |
|---|---|
| | <ul> <li>Subjects will come back for a 4-week posttreatment follow up visit at Week 12 (Day 84).</li> <li>Participant's safety will be monitored throughout the study. Safety will be assessed by monitoring reported adverse events, vital signs, clinical chemistry and hematology and overall tolerability of the investigational product.</li> <li>Subjects would be required to discontinue the investigational product under the following circumstances: <ul> <li>Development of an intercurrent illness that would jeopardize the safety, or significantly affect assessments of clinical status of a subject</li> <li>Either at the discretion of the Investigator or at the participant's request</li> <li>Development of any investigational product-related SAE</li> <li>Suspected or laboratory-confirmed pregnancy</li> </ul> </li> </ul> |
| Number of<br>Subjects and Sites | Approximately 130 subjects are planned to be enrolled, and assuming a 20% drop out rate, the planned overall sample size for this clinical trial is approximately 104 adult male and female subjects, 18 years of age and older with mild to moderate rosacea. Subjects will be randomized at a 1:1 ratio (B244: vehicle) at about 8 clinical research centers in the United States. |
| | INCLUSION CRITERIA |
| Eligibility Criteria | <ul> <li>Male a n d f e male subjects 18.</li> <li>A clinical diagnosis of mild to moderate facial rosacea.</li> <li>In good general health as determined by a thorough medical history, physical examination, clinical chemistry and hematology.</li> <li>A Clinician Erythema Assessment (CEA) score of 2-3 at Screening and at Baseline Visits (prior to the investigational product application).</li> <li>Mild to Moderate IGA score of 2-3 at Screening and at Baseline Visits (prior to the investigational product application).</li> </ul> |
| | <ul> <li>Willing to refrain from using any topical or systemic treatments for the treatment of rosacea, other than the investigational product.</li> <li>Females of childbearing potential with a negative urine pregnancy test (UPT) at Screening and Baseline/Day 1 (prior to the investigational product application).</li> <li>Ability to comprehend and comply with study procedures.</li> <li>Agree to commit to participate in the current protocol.</li> </ul> |

STATISTICAL ANALYSIS PLAN





 Provide written informed consent prior to any study procedure being performed.

#### **EXCLUSION CRITERIA**

Any subject who meet one or more of the following criteria are excluded from this study.

- Female subjects who are pregnant, lactating or who are trying to conceive will be excluded from participation in this study.
- Any uncontrolled chronic or serious disease or medical condition that would normally prevent participation in a clinical trial, or, in the judgment of the Investigator, would put the subject at undue risk, or might confound the study assessments (e.g., other dermatological diseases), or might interfere with the subject's participation in the study, (e.g., planned hospitalization during the study).
- Particular forms of rosacea (e.g., rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin, Ocular rosacea Phymatous rosacea, Steroid-induced rosacea, severe rosacea including pyoderma faciale) or other concomitant facial dermatoses that are similar to rosacea such as peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus, or actinic telangiectasia.
- Presence of three (3) or more facial inflammatory lesions of rosacea
- Any skin condition which in the investigator's opinion may interfere with the evaluation of rosacea.
- Severe papulopustular rosacea requiring systemic treatment.
- Participation at the time of eligibility assessment (Screening) in any other investigational drug or device study or may have participated within 30 days prior to Screening.
- Commencement of new hormonal therapy or dose change to hormonal therapy within 90 days prior to baseline. Dose and frequency of use of any hormonal therapy started more than 90 days prior to baseline must remain unchanged throughout the study. Hormonal therapies include, but are not limited to, oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (e.g. vaginal ring or transdermal hormone contraception).





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN Version 1

- Presence of beard or excessive facial hair at Screening which would interfere with the study treatments or study assessments and refusal to remove for duration of study.
- Current treatment with monoamine oxidase (MAO) inhibitors, barbiturates, opiates, sedatives, systemic anesthetics, or alphaagonists.
- Carcinoid, Pheochromocytoma or other systemic causes of flushing.
- Known sensitivity to B244 or its components.
- Refusal to submit to blood and urine sampling for laboratory analysis.
- Treatment with the following:

**Prohibited Topical Treatments:** 

| Pronibited Topical Treatments: | |
|---|---|
| Topical Treatment | Prohibited Time<br>Frame prior to<br>Baseline |
| Astringents or abrasives | 2 days |
| RHOFADE™ (oxymetazoline HCl) Cream,1% | 1 week |
| Bleach baths | 1 week |
| Mirvaso (brimonidine) topical cream | 1 week |
| Vinegar | 1 week |
| Topical Prescription/OTC medications for | 1 week |
| treatment of acne | |
| Soolantra (Ivermectin 1%) topical cream | 1 week |
| Topical Antibiotic | 2 weeks |
| Use of over the counter antimicrobial | 2 weeks |
| Benzoyl Peroxide | 2 weeks |
| Immunomodulators | 4 weeks |
| Oracea (doxycycline) topical cream | 2 weeks |
| Corticosteroids | 4 weeks |
| Electrocoagulation, Dermabrasion; Facial | 4 weeks |
| peels | 4 1 |
| Dermatologic/surgical procedure on the face | 4 weeks |
| | 4 weeks |
| Topical Prescription medications for the | 4 weeks |
| treatment of rosacea (e.g. azelaic acid, metronidazole, etc.) | |
| , , | 4 weeks |
| Laser, Phototherapy, Photodynamic | 4 weeks |
| Therapy or IPL (intense pulsed light) | |
| treatment | |





|---|---|---|
| | Prescription or over the counter topical retinoid use on the face (e.g., tretinoin, tazarotene, adapalene) | 4 weeks |
| | Prohibited Systemic Treatments: | |
| | Topical Treatment | Prohibited Time Frame prior to Baseline |
| | Exposed to excessive ultraviolet (UV) radiation and/or subject was unwilling to refrain from excessive exposure to UV radiation during the course of the study. | 1 week |
| | Prescription anti inflammatory Prescription/OTC anti-inflammatory | 2 weeks<br>2 weeks |
| | medications (excludes low dose aspirin) Systemic Antibiotics | 4 weeks |
| | Prescription medications for the treatment of rosacea (e.g. doxycycline, tetracycline, macrolides) | 4 weeks |
| | Prescription medications for treatment of acne | 4 weeks |
| | Corticosteroids (oral or injectable) | 4 weeks |
| | Immunomodulators Oral retinoid use (e.g., isotretinoin), vitamin A supplements greater than 10,000 units/day | 12 weeks 6 months |
| Withdrawal and<br>Early<br>Discontinuation | drawal and A subject may voluntarily withdraw from the study at any time and for any reason without prejudice to his or her future medical care. The Investigator Sponsor or Medical Monitor may also withdraw a subject | |
| Prohibited<br>Concomitant<br>Medication | methods that are not allowed during the study period and within the | |
| Study Drug | supply study drug as matching 30mi/bottle, labeled for a billided study. | |
| | <ul> <li>Test Drug: B244, 30ml/bottle (AOBion</li> <li>Placebo: Vehicle, 30ml/bottle (AOBion</li> </ul> | |





|---|---|
| Duration of Patient<br>Study Participation | Up to $84 \pm 2$ days |
| Study Endpoints | PRIMARY |
| | • The primary safety endpoint is to assess the safety and tolerability of B244 applied twice daily (BID) to the face for 8 weeks in subjects with mild to moderate rosacea based on the number of AE & SAE. |
| | EXPLORATORY |
| | To assess the efficacy of B244 in subjects with mild to moderate rosacea. |
| | <ul> <li>Change of IGA score at Baseline to Week 1, Week 4, Week 8<br/>and Week 12</li> </ul> |
| | <ul> <li>Change of CEA score at Baseline to Week 1, Week 4, Week 8<br/>and Week 12.</li> </ul> |
| | <ul> <li>Change of PSA score at Baseline to Week 1, Week 4, Week 8 and Week 12.</li> <li>Change of Skindex 16 patient reported outcome from Baseline to Week 1, Week 4, Week 8 and Week 12</li> </ul> |
| | • IGA treatment success, defined as "clear" or "almost clear" with a 2-grade improvement in IGA score from baseline to the end of treatment. |
| | • CEA treatment success, defined as "clear" or "almost clear" with a 2-grade improvement in CEA score from baseline to the end of treatment |
| Statistical Analysis | SAFETY ANALYSIS |
| | The reporting of safety data is descriptive (arithmetic mean, standard deviation (SD), coefficient of variation (CV), median, minimum, and maximum) will be calculated for quantitative safety data as well as for the difference from baseline, when appropriate. |
| | The analysis will include all subjects who receive at least one dose of investigational product. The variables for safety endpoints are AEs, Local Application Site Reactions, vital signs measurements, clinical chemistry and hematology. AEs will be summarized based on the frequency of AEs and their severity for all treated subjects. All AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA) and summarized by treatment group. Data will be summarized using preferred term and primary system organ class, including verbatim term, dose level, severity, and relationship to treatment, will be provided. |






Concomitant medications will be listed by treatment and coded using the most recent version of the World Health Organization (WHO) Drug Dictionary (DD).

# **EFFICACY ANALYSIS**

The Evaluable Period for the outcome variables will be weeks 1, 4, 8 and 12. The superiority of the drug over the vehicle will be tested at week 8 based on the probability of improvement from baseline with a continuity-corrected Z-tests comparing the change from baseline of treatments vs Placebo. For all other evaluable periods, descriptive statistics for the change from baseline will be shown.

The change from baseline score of Skindex-16 will be compared among treatments at Week 12 using an ANOVA.






# STATISTICAL ANALYSIS PLAN


# **Table of Contents**

# Contents

| S | ΓATIS | ΓΙCAL ANALYSIS PLAN REVIEW AND APPROVAL | 2 |
|---|---|---|---|
| ΡF | котос | OL SYNOPSIS | 3 |
| 1 | LIST | OF ABBREVIATION | 14 |
| 2 | INT | RODUCTION | 16 |
| | 2.1 | Study Overview | 16 |
| | 2.2 | Study Flowchart | 18 |
| | 2.3 | Schedule of Activities | 19 |
| 3 | STU | DY OBJECTIVE AND ENDPOINTS | 21 |
| | 3.1 | Study Objectives | 21 |
| | 3.1. | 1 Primary Objective | 21 |
| | 3.1. | 2 Exploratory Objectives | 21 |
| | 3.2 | Study Endpoints | 21 |
| | 3.2. | 1 Safety & Tolerability (Primary) | 21 |
| | 3.2. | 2 Efficacy (Exploratory) | 21 |
| 4 | STU | DY DESIGN | 22 |
| | 4.1 | Summary of Study Design | 22 |
| | 4.2 | Definition of Study Drugs | 22 |
| | 4.3 | Sample Size Considerations | 23 |
| | 4.4 | Study Withdrawal | 23 |
| | 4.5 | Early Discontinuation | 24 |
| 5 | PLA | NNED ANALYSIS | 24 |
| | 5.1 | Final Analysis | 24 |
| 6 | GEN | IERAL CONSIDERATION FOR DATA ANALYSIS AND HANDLING | 24 |
| | 6.1 | General Summary Table and Individual Subject Data Listing | 24 |
| | 6.2 | General Summary Table and Individual Subject Data Listing Considerations | 25 |
| | 6.3 | Data Management | 26 |
| | 6.4 | Data Presentation Conventions | 26 |
| | 6.5 | Analysis Populations | 27 |
| | 6.5. | 1 Screen Failures | 27 |





| Protocol: RE Confidential | | Version 1<br>14-Feb-19 |
|---|---|---|
| 6.5.2 | Safety Population | |
| 6.5.3 | mITT Population | 27 |
| 6.5.4 | Per-Protocol (PP) Population | 27 |
| 6.6 Ba | seline Definition | 28 |
| 6.7 De | rived and Transformed Data | 28 |
| 6.7.1 | Baseline Age | 28 |
| 6.7.2 | Study Day | 28 |
| 6.7.3 | Multiple Assessments | 28 |
| 6.7.4 | Handling of Missing Data & Sensitivity Analysis | 28 |
| 6.7.5 | Missing Start and Stop Dates for Prior and Concomitant Medication | 29 |
| 6.7.6 | Safety Parameters | 29 |
| 6.7.7 | Missing Start and Stop Dates for Adverse Events | 29 |
| 7 DATA A | NALYSES | 31 |
| 7.1 Su | bjects Disposition | 31 |
| 7.2 Pr | otocol Deviations | 31 |
| 7.3 De | mographic and Baseline Characteristics | 32 |
| 7.4 St | udy Drug Exposure | 32 |
| 7.5 M | edical History | 32 |
| 7.6 Co | ncomitant Medication | 33 |
| 7.7 Vit | al Signs and Physical Examination | 33 |
| 7.8 La | boratory Data | 33 |
| 7.9 Vis | sit Windows | 33 |
| 8 STATIST | ΓΙCAL ANALYSES | 33 |
| 8.1 Sa | mple Size Determination | 33 |
| 8.2 Sa | fety Analysis | 34 |
| 8.2.1 | Primary Safety Endpoint | 34 |
| 8.3 Eff | icacy Analysis | 34 |
| 8.4 Se | nsitivity Analysis | 35 |
| 9 REFERE | NCES | 36 |
| 10 APPE | NDIX | 37 |
| 10.1 AP | PENDIX A: Tables | 37 |
| 10.1.1 | General | 37 |





| Protocol: RB2 | 44-001 STATISTICAL ANALYSIS PLAN | Version 1 |
|---------------|----------------------------------|-----------|
| 10.1.2 | Efficacy | 49 |
| | Safety | |
| | ENDIX B: Listings | |
| 10.2 APP | ENDIX B. LISTINGS | |
| 10 2 ADD | FNDIX C. Figures | 5.0 |



Protocol: RB244-001 STATISTICAL ANALYSIS PLAN Version 1 Confidential 14-Feb-19

# 1 LIST OF ABBREVIATION

| Abbreviation | Full Form |
|--------------|------------------------------------------------|
| AE | Adverse Event |
| AOB | Ammonia-Oxidizing Bacteria |
| BID | Bis in Die (twice a day) |
| BP | Blood Pressure |
| CEA | Clinician Erythema Assessment |
| CRA | Clinical Research Associate |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CTMF | Clinical Trial Master File |
| CTP | Clinical Trial Protocol |
| eCRF | Electronic Case Report Form |
| EOS | End of Study |
| ET | Early Termination |
| ETR | Erythematotelangiectatic rosacea |
| GCP | Good Clinical Practice |
| IB | Investigator's Brochure |
| ICH | International Conference On Harmonization |
| IEC | Independent Ethics Committee |
| IGA | Investigator Global Assessment |
| IGE | Investigator's Global Evaluation |
| IP | Investigational Product |
| IPL | Intense Pulsed Light |
| IRB | Institutional Review Board |
| ISF | Investigator Site File |
| IUD | Intrauterine Device |
| IUS | Intrauterine system |
| IWRS | Interactive Web Response System |
| LOCF | Last Observation Carried Forward |
| mITT | Modified Intent-To-Treat |
| NSAID | Nonsteroidal Anti-inflammatory Drug |
| OTC | Over the Counter |
| PP | Per-Protocol |
| PRN | Pro Re Nada (as needed) |
| PRN | Pro Re Nada (as needed) |
| PSA | Patient Self-Assessment |
| RR | Relative Risk |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SI | Simple Imputation |
| SOP | Standard Operating Procedures |
| SUSAR | Suspected Unexpected Serious Adverse Reactions |
| TEAE | Treatment Emergent Adverse Event |
| | _ |





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN Version 1 Confidential 14-Feb-19

Upper Limit of Normal Range Urine Pregnancy Test Ultraviolet ULN

UPT

UV

White Blood Cell Count WBC





# 2 INTRODUCTION

This document describes the statistical methods and data presentations to be used in the summary and analysis of data from Protocol RB244-001. Background information is provided for the overall study design and objectives. The reader is referred to the study protocol and electronic case report forms (eCRFs) for details of study conduct and data collection.

# 2.1 Study Overview

The proposed study is aimed to evaluate the safety and efficacy of B244 topical spray. A Vehicle-Controlled, Double-Blind, Multicenter, Randomized Study Design has been Selected to Evaluate the Safety and Efficacy of the B244 Investigational product in the Treatment of Mild-to-Moderate Rosacea.

There is no cure for rosacea and treatment is aimed at alleviating the symptoms. Topical or oral medications are generally prescribed for mild to moderate papulopustular rosacea. These topical medications include: metronidazole, azelaic acid, sodium sulfacetamide and sulfur, erythromycin, and tretinoin8. Currently these approved topical medications may cause local irritation to the skin. The oral medications prescribed for severe disease include tetracycline, doxycycline, minocycline, erythromycin and metronidazole. The systemic therapies may result in systemic adverse events such as gastrointestinal upset and photosensitivity.

It is believed, that topical application of Ammonia-Oxidizing Bacteria (AOB) will reduce survival of pathogenic bacteria present on the skin and thus improve rosacea symptoms in those affected by it. B244 is being developed as a 'live topical' to provide a natural source of AOB and NO/NO2 to the human skin.

This is a Prospective, Vehicle Controlled, Double Blind, Multicenter, Randomized Phase II trial, Comparing the effect of twice daily B244 application for 8 weeks vs. vehicle application on treatment of mild to moderate rosacea. At Screening and Baseline all subjects must have clinical diagnosis of mild to moderate rosacea and subjects must have IGA score of 2-3 and CEA score of 2-3 to qualify for the study.

After screening and recruitment, participants will be randomized to active or vehicle application for 8 weeks. Subjects will apply a total of 4 pumps of IP per application to the face twice-a-day. Subjects will be provided with cleanser and moisturizer to use for the duration of the study. All B244 randomized subjects will be treated at the dose of  $4 \times 10^9$  cells/ml via spray application.

Efficacy will be assessed using Investigator Global Assessment (IGA) score, Clinician's Erythema Assessment (CEA) score, Patient Self-Assessment (PSA) score and patient reported Skindex 16. Participant's safety will be monitored throughout the study. Safety



# AOBiome

Version 1

14-Feb-19

# CLINICAL RESEARCH OPTIMIZED™

Protocol: RB244-001 STATISTICAL ANALYSIS PLAN

will be assessed by monitoring reported adverse events, vital signs, clinical chemistry and hematology and overall tolerability of the investigational product.

Approximately 130 subjects are planned to be enrolled, and assuming a 20% drop out rate, the planned overall sample size for this clinical trial is approximately 104 adult male and female subjects, 18 years of age and older with mild to moderate rosacea. Subjects will be randomized at a 1:1 ratio (B244: Vehicle) at about 8 clinical research centers in the United States.

The entire study will consist of a total of 6 visits:

- Visit 1(Day -21 to -1): Screening will occur at Days -21 to -1, followed by Washout (Days -14 to -1).
- Visit 2(Baseline/ Day 1): Randomization will occur during the baseline visit for the study (Day 1).
- Visit 3 5(Day 7 ± 2 [Week 1], Day 28 ± 2 [Week 4], Day 56 ± 2 [Week 8]): Clinical assessments of response to treatment will be made at Week 1(Day 7), Week 4 (Day 28), and Week 8 (Day 56).
- Visit 6(Day  $84 \pm 2$ ): Subjects will come back for a 4-week post-treatment follow up visit at Week 12 (Day 84).





STATISTICAL ANALYSIS PLAN Protocol: RB244-001


#### 2.2 **Study Flowchart**

Figure 1. Study Flowchart

# STUDY SCHEMA







Protocol: RB244-001 STATISTICAL ANALYSIS PLAN


#### **Schedule of Activities** 2.3

CLINICAL RESEARCH OPTIMIZED™

 Table 1: Schedule of Study Activities

| Visit Name | Screening | Baseline/ DAY 1 | Week<br>1 | Week 4 | Week 8 | Week 12/<br>End of<br>Study Visit | Early<br>Termination<br>Visit |
|---|---|---|---|---|---|---|---|
| Visit number | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | |
| Visit window in days | -21 to -1 | 1 | 7+/-2 | 28 +/- 2 | 56 +/- 2 | 84 +/- 2 | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | X | | | | | |
| Demographics | X | | | | | | |
| Medical History | X | X | | | | | |
| Concomitant Medications | X | X | X | X | X | X | X |
| Physical Exam | X | X | | | | X | X |
| BP & Pulse <sup>2</sup> | X | X | X | X | X | X | X |
| Urine pregnancy test for WOCBP <sup>1</sup> | X | X | X | X | X | X | X |
| Clinical chemistry and hematology and urinalysis <sup>3</sup> | X | X | | X | X | | X |
| Biomarkers <sup>4</sup> | | X | | | X | | X |
| CEA | X | X | X | X | X | X | X |
| IGA | X | X | X | X | X | X | X |
| Skindex 16 | X | X | X | X | X | X | X |
| PSA score | X | X | X | X | X | X | X |
| Telangiectasia Evaluation | | X | | | X | | X |
| Fitzpatrick skin type | X | | | | | | |
| IWRS | | X | | X | | | |
| Dispense Investigational product to Subject 5/6 | | X | | X | | | |
| Collect Investigational product from Subject <sup>5</sup> | | | | X | X | | X |





#### 1 DDA44 001 CTATICTICAL ANALYCIC DLAN


| Visit Name | Screening | Baseline/<br>DAY 1 | Week<br>1 | Week 4 | Week 8 | Week 12/<br>End of<br>Study Visit | Early<br>Termination<br>Visit |
|---|---|---|---|---|---|---|---|
| Visit number | Visit 1 | Visit 2 | Visit<br>3 | Visit 4 | Visit 5 | Visit 6 | |
| Visit window in days | -21 to -1 | 1 | 7+/-2 | 28 +/- 2 | 56 +/- 2 | 84 +/- 2 | |
| Investigational product<br>Compliance <sup>5</sup> | | X | | X | X | | X |
| Study Cleanser and moisturizer dispensation <sup>9</sup> | | X | | X | | | |
| Study Cleanser and moisturizer collection | | | | | X | | X |
| Study Diary <sup>8</sup> | | X | X | X | X | | X |
| Study Counseling <sup>7</sup> | | X | X | X | X | | |
| AE Collection and<br>Assessment | X | X | X | X | X | X | X |

- 1. Urine pregnancy test for WOCBP will be done at every visit.
- 2. Blood pressure readings will be obtained at every visit. Subject should be allowed to rest for more than 5 minutes sitting, then BP measurements and pulse (x3) will be performed, using the non-dominant arm with a calibrated electronic sphygmomanometer. The average of the second and third readings will be documented.
- 3. Subjects should fast for at least 8 hours before the test. Laboratory work includes: hematology and Lipid Panel, Albumin, Alkaline Phos, ALT, AST, Total Bilirubin, BUN, BUN: Creatinine ratio, Calcium, Chloride, Creatinine, eGFR, Glucose, Potassium, Sodium, Uric Acid, and urinalysis. HIV Ab, HCV Ab, HBsAg. will only be done at screening.
- 4. Subjects should fast for at least 8 hours before the test.
- 5. Weight of the investigational product kit will be obtained at the Baseline visit. Study staff will be asked to weigh all dispensed bottles without the carton box PRE- FIRST DOSE. Weight will be recorded in grams.
- 6. Subjects will be asked to bring all dispensed bottles back for the Week 4 and Week 8 visits. Upon return for the study visit, all bottles will be weighed again without the carton box. Subjects will be asked to apply the investigational product twice daily. First investigational product application will happen at the site under medical supervision.
- 7. Subjects will be counseled on the use of study medication and answer any questions subject may have.
- 8. Subjects will be asked to fill out study diary for the duration of the study.
- 9. Cleanser and moisturizer will be dispensed at the Baseline visit. Subjects will be asked to refrain, if possible, from using any other cleanser and/or moisturizer on their face and apply the provided product while they are participating in the trial. Any leftover moisturizer /cleanser will be collected at Week 8 visit, at which point subjects will be asked to go back to their regular routine.





# 3 STUDY OBJECTIVE AND ENDPOINTS

# 3.1 Study Objectives

# 3.1.1 Primary Objective

To assess the safety and tolerability of B244 applied twice daily (BID) to the face for 8 weeks in subjects with mild to moderate rosacea.

# 3.1.2 Exploratory Objectives

To assess the efficacy of B244 in subjects with mild to moderate rosacea.

- o Proportion of subjects with IGA improvement at Week 8 relative to baseline.
- o Proportion of subjects with CEA improvement at Week 8 relative to baseline.
- o Change in IGA from Week 8 to Baseline.
- o Change in CEA from Week 8 to Baseline.
- o Proportion of Subjects with improvement in IGA or CEA at Week 1, Week 4, and Week 12.
- Change in Skindex 16 patient reported outcome from Baseline to Week 1, Week 4, Week 8, and Week 12.
- o Proportion of subjects with change in PSA at Week 1, Week 4, Week 8 and Week 12 from Baseline.
- Evaluation of Telangiectasia Score at Baseline/Day 1 and Week 8

# 3.2 Study Endpoints

# 3.2.1 Safety & Tolerability (Primary)

Safety and tolerability endpoints will consist of all adverse events reported during the study duration.

# 3.2.2 Efficacy (Exploratory)

- o Change of IGA score at Baseline to Week 1, Week 4, Week 8 and Week 12.
- o Change of CEA score at Baseline to Week 1, Week 4, Week 8 and Week 12.
- o Change of PSA score at Baseline to Week 1, Week 4, Week 8 and Week 12.
- Change of Skindex 16 patient reported outcome from Baseline to Week 1, Week 4, Week 8 and Week 12.
- o IGA treatment success, defined as "clear" or "almost clear" with a 2-grade improvement in IGA score from baseline to the end of treatment.
- o CEA treatment success, defined as "clear" or "almost clear" with a 2-grade improvement in CEA score from baseline to the end of treatment.





# 4 STUDY DESIGN

# 4.1 Summary of Study Design

This is a Prospective, Vehicle Controlled, Double Blind, Multicenter, Randomized Phase II trial, Comparing the effect of twice daily B244 application for 8 weeks vs. vehicle application on treatment of mild to moderate rosacea. We will enroll approximately 130 subjects and complete 104 subjects.

At Screening and Baseline, all subjects must have clinical diagnosis of mild to moderate rosacea and must have IGA score of 2-3 and CEA score of 2-3 to qualify for the study. After screening and recruitment, participants will be randomized to active or vehicle application for 8 weeks. Subjects will apply a total of 4 pumps of IP per application to the face twice-a-day. Randomization will be 1:1 B244 to Vehicle. Subjects will be provided with cleanser and moisturizer to use for the duration of the study. All B244 randomized subjects will be treated at the dose of  $4x10^9$  cells/ml via spray application. Screening will occur at Days -21 to -1. Washout will occur after Screening visit (Days -14 to -1) and randomization will occur during the baseline visit for the study (Day 1).

Efficacy will be assessed using Investigator Global Assessment (IGA) score, Clinician's Erythema Assessment (CEA) score, Patient Self-Assessment (PSA) score and patient reported Skindex 16. Clinical assessments of response to treatment will be made at Week 1(Day 7), Week 4 (Day 28), and Week 8 (Day 56). At Baseline visit, subjects will receive a kit containing the drug product. Each bottle will be used for 2 weeks. At Week 4, subjects will return the used bottles from the kit and will be issued a new kit of drug product to be used from Week 4 through Week 8. Subjects will stop applying investigational product at Week 8 and will return investigational product at that visit. Subjects will come back for a 4-week post-treatment follow up visit at Week 12 (Day 84). Participant's safety will be monitored throughout the study. Safety will be assessed by monitoring reported adverse events, vital signs, clinical chemistry and hematology and overall tolerability of the investigational product.

Subjects would be required to discontinue the investigational product under the following circumstances:

- Development of an intercurrent illness that would jeopardize the safety, or significantly affect assessments of clinical status of a subject
- Either at the discretion of the Investigator or at the participant's request
- Development of any investigational product-related SAE
- Suspected or laboratory-confirmed pregnancy

# 4.2 Definition of Study Drugs

Study drug includes Test and Placebo drug products. The Sponsor will supply study drug as matching 30ml/bottle, labeled for a blinded study.






Test Drug: B244, 30ml/bottle (AOBiome, LLC)
Placebo: Vehicle, 30ml/bottle (AOBiome, LLC)

# 4.3 Sample Size Considerations

Approximately 130 subjects are planned to be enrolled, and assuming a 20% drop out rate, the planned overall sample size for this clinical trial is approximately 104 adult male and female subjects, 18 years of age and older with mild to moderate rosacea. Subjects will be randomized at a 1:1 ratio (B244: Vehicle) at about 9 clinical research centers in the United States.

# 4.4 Study Withdrawal

A subject may voluntarily withdraw from the study at any time and for any reason without prejudice to his or her future medical care. The Investigator, Sponsor, or Medical Monitor may also withdraw a subject at any time if it is medically necessary or in the interest of subject's safety. Additional reasons for premature discontinuation of investigational product may include adverse events and major non-compliance with study procedures, as described below. The withdrawal of a subject from investigational product by the Investigator will be discussed with the Medical Monitor before the subject stops investigational product, whenever possible.

A subject will be discontinued from this study if any of the following criteria are met:

- Withdrawal of consent by the subject is received.
- In the opinion of the Investigator, Medical Monitor or Sponsor, it is not in the subject's best interests to continue in the study.
- Significant non-compliance with study procedures that would interfere with the study results or increase the subject's risks in the study, as determined by the Investigator.
- Development of an intercurrent illness that would jeopardize the safety, or significantly affect assessments of clinical status of a subject.
- Development of any investigational product-related SAE.
- Suspected or laboratory-confirmed pregnancy.

Subjects who discontinued early from the study due to lack of treatment effect after completing at least four weeks of treatment (Day 28) will be included in the mITT and PP population as treatment failures and the change in IGA and CEA from the baseline visit to the last completed visit prior to discontinuation due to lack of efficacy will be carried forward in the primary endpoint analysis. Subjects discontinued early for other reasons will be excluded from the PP population.





# 4.5 Early Discontinuation

CLINICAL RESEARCH OPTIMIZED™

If a subject discontinues prematurely, the Investigator will perform Early Termination (ET) visit, capturing the reason for discontinuation.

If a subject does not return for a scheduled visit, every effort will be made to contact the subject and document the End of Study visit assessments. The Investigator must document the primary reason for discontinuation of a study subject in the source document and on the appropriate electronic case report form (eCRF).

# 5 PLANNED ANALYSIS

# 5.1 Final Analysis

Final analysis is planned for the study after the database lock. The final analysis will follow instructions presented in this SAP.

# 6 GENERAL CONSIDERATION FOR DATA ANALYSIS AND HANDLING

# 6.1 General Summary Table and Individual Subject Data Listing

Summary tables and listings (e.g., post text tables and individual subject data listings are prepared according to ICH Guideline E3) include a "footer" providing explanatory notes that indicate as a minimum:

- SAS program name.
- Programmer.
- Date of data extraction.
- Date of output generation.

Post text tables also include reference(s) to the subject data listing(s) that supports the summary data. The data extraction date links the output to the archived database that is locked to ensure the replication of the results.

Post text tables will be organized with respect to treatment group and a column will be included to summarize all treated subjects. The order of drug presentation will be investigational drug first followed by the vehicle control. A total column will appear as the last column. The summary tables clearly indicate the number of subjects to which the data apply and unknown or not performed are distinguished from missing data.

Summary tables for medications and medical conditions are coded according the WHO Drug Dictionary. Adverse event preferred terms and body/organ systems are coded using





Version 1

Protocol: RB244-001 STATISTICAL ANALYSIS PLAN


the MedDRA dictionary. The MedDRA dictionary can be used, as well, in the coding of signs and symptoms, medical history, physical examination abnormalities, and clinical diagnoses.

Supportive individual subject data listings, as a minimum, are sorted and presented by treatment group and subject id. Listings also include visit number, visit date, and days relative to the initiation of double-blind treatment.

# 6.2 General Summary Table and Individual Subject Data Listing Considerations

The default convention is to number tables and listings using a decimal system to reflect main levels of unique tables and listings and sub-levels of replicate tables and listings with two digits per level (e.g., Table XX.YY.ZZ. ...).

- The first level number should be consistent with the corresponding CSR appendix in which the tables or listings will appear. For example, the post text tables usually occupy Appendix 14 and the individual subject data listings are put in Appendix 16. All post text tables should have a main number level 14 and listings 16. The subject accounting and disposition table is usually first in the first section of the report and should be numbered Table 14.1. The supportive subject data listing would be Listing 16.1. A subset by sex 2. Subject accounting and final disposition should appear as the second level number (Table 14.1 series). Baseline and demographic profile occupy the next sub-level (Table 14.2 series). Efficacy should come next (Table 14.3 series) followed by safety Table 14.4 series). Reasons for subjects' being excluded from efficacy and protocol violation summary tables should appear as the last level (Table 14.5 series). Similar conventions should be applied to the subject data listings.
- The title should be complete, accurate, and concise. The last line of the title should provide the analysis group being summarized (e.g., Intent-to-Treat Subjects or Per-Protocol Efficacy Subjects). If possible, the units of measurement for data contained in the table can appear in parentheses to conserve space in the body of the table. For example, the summary of vital signs title could read "Summary of Sitting and Standing Blood Pressure (mmHg) and Heart Rate (bpm)." Whether in the title or body of a table or listing, units must always be specified for all appropriate data.
- If possible, variables being summarized, and statistics reported should appear in the left most column of a table. The next columns for treatment groups should report the data from left to right for the investigational drug, placebo, comparative agents, and (optional) all treated subjects, respectively.

In general, the listings should be sorted and presented by treatment assignment, investigational site, and subject number. Treatment assignment and site can appear in the banner of the listing. From left to right, the subject number, visit number, visit date, and relative day should appear.





Version 1

Protocol: RB244-001 STATISTICAL ANALYSIS PLAN


All tables and listings must have explanatory notes that give, as a minimum, data extraction date, output generation date, complete program name and path where it is stored, as appropriate. The definition of all derived variables and decodes for coded data must appear in the notes. Due to space limitations, tables and listings may require a page of notes as a one-time preface to the output.

# 6.3 Data Management

Biorasi will create SDTM data sets and ADaM analysis data sets using (SAS®) software. Data analyses and summary tables are generated using SAS version 9.4 or above

#### **6.4 Data Presentation Conventions**

Continuous variables (e.g. age) are summarized using descriptive statistics (the number of subjects with available data, the mean, standard deviation (SD), median, minimum and maximum). Categorical variables (e.g. race) are summarized using counts and percentages. Percentages are calculated using the total subjects per treatment group.

The following conventions are applied to all data presentations and summaries:

- For continuous variables, all mean and median values are formatted to one more decimal place than the measured value. Standard deviation values are formatted to two more decimal places than the measured value. Minimum and maximum values are presented with the same number of decimal places as the measured value.
- For categorical variables, the number and percentage of responses are presented in the form XX (XX.X %) where the percentage is in the parentheses.
- Date variables are formatted as DDMMMYYYY for presentation. Time is formatted in military time as HH:MM for presentation.
- Wherever possible, data will be decimal aligned.
- P-values, if applicable, will be presented to 4 decimal places. If the p-value is less than 0.0001 then it will be presented as <0.0001.

Unless otherwise stated, any statistical tests performed will use 2-sided tests at the 5% significance level.

The table and listing shells and table of contents as part of this SAP provide the expected layout and titles of the tables, listings and figures. Any changes to format, layout, titles, numbering, or any other minor deviation will not necessitate a revision to the SAP nor will it be considered a deviation from planned analyses. Only true differences in the analysis methods or data handling will necessitate such documentation. The appropriate listings supporting the tables will be included and are not specified in the individual sections throughout the document.





# 6.5 Analysis Populations

#### 6.5.1 Screen Failures

Investigators must account for all subjects who sign informed consent and will maintain an Enrollment Log capturing subjects screened and indicating who was enrolled or excluded and the reason why. If the subject is found not to be eligible prior to enrollment, the reason(s) for ineligibility must be documented by the Investigator.

These subjects will neither contribute to data presentations nor be included in formal statistical analyses. The number of screen failures will be included in the data disposition table. Subject Numbers assigned to subjects who fail Screening will not be re-used.

# **6.5.2 Safety Population**

The safety population includes all randomized subjects who received investigational product.

## 6.5.3 mITT Population

A modified intent-to-treat population includes all subjects who are randomized, applied at least one dose of assigned product, and returned for at least one post-baseline evaluation visit.

# 6.5.4 Per-Protocol (PP) Population

The PP population includes all randomized subjects who met all inclusion/exclusion criteria, were compliant with the assigned study treatment, returned to the study site for the primary endpoint visit within the specified window ( $\pm 2$  days) OR discontinued from the study as a treatment failure, and did not have any major protocol violations.

Subjects who administered at least 50 % of IP, have at least one baseline and post baseline in clinic visit and did not have any major protocol violations.

Subjects who discontinued early from the study due to lack of treatment effect after completing at least eight weeks of treatment should be included in the mITT and PP population as treatment failures and the change in IGA and CEA from the baseline visit to the last completed visit prior to discontinuation due to lack of efficacy should be carried forward in the primary endpoint analysis. Subjects discontinued early for other reasons should be excluded from the PP population but included in the mITT population.

The results in the mITT population will be considered definitive for superiority of each active treatment to vehicle with those in the PP population considered supportive. Safety analyses will be performed using the Safety population.



Protocol: RB244-001 STATISTICAL ANALYSIS PLAN


#### 6.6 **Baseline Definition**

CLINICAL RESEARCH OPTIMIZED™

The Baseline visit (Day 0) will take place once the results of Screening assessments are obtained, suggesting that the subject is eligible for entering the study. During this visit, those subjects who qualify for entering the study will be randomized to one of the study arms in a ratio of 1:1.

#### **6.7 Derived and Transformed Data**

### 6.7.1 Baseline Age

Subject's age in years will be calculated based on the date of the Baseline Visit date using the following formula:

Age (years) = FLOOR ((INTCK ('month', Date of Birth, Date of Baseline Visit) -(DAY(Date of Baseline Visit) < MIN(DAY(Date of Birth), DAY (INTNX ('month', Date of Baseline Visit, (1) - (1) / (12); where:

- o FLOOR () is a SAS function that returns the largest integer that is less than or equal to the argument.
- o INTCK () is a SAS function that returns the number of interval boundaries of a given kind that lie between two dates, times, or datetime values.
- DAY () is a SAS function that returns the day of the month from a SAS date value.
- INTNX () is a SAS function that increments a date, time, or datetime value by a given time interval, and returns a date, time, or datetime value.

## 6.7.2 Study Day

Day 1 is defined as the day after the baseline when the subject will receive the first dose.

- o For a visit date on or after the date of the first dose: Study Day = (date of interest - date of first dose) + 1
- o For a visit date before the date of the first dose: Study Day = (date of interest - date of first dose)

# **6.7.3** Multiple Assessments

No multiple assessment for same visit are scheduled.

## 6.7.4 Handling of Missing Data & Sensitivity Analysis

For the primary and secondary analysis no missing values will be imputed. A sensitivity analysis will be performed by Multiple Imputation Regression Analysis using the following factors: treatment, age, gender, race, baseline IGA, baseline CEA, baseline PSA, smokers/non-smokers and the results of the same variable from previous visits.





STATISTICAL ANALYSIS PLAN

Protocol: RB244-001 Version 1 Confidential 14-Feb-19

# 6.7.5 Missing Start and Stop Dates for Prior and Concomitant Medication

#### Start date:

- o If start date is completely missing, start date will not be imputed.
- o If (year is present, and month and day are missing) or (year and day are present, and month is missing), set month and day to January 1.
- o If year and month are present and day is missing, set day to the 1st day of month

# Stop date:

- o If end date is completely missing, end date will not be imputed.
- o If (year is present, and month and day are missing) or (year and day are present, and month is missing), set month and day to December 31st.
- o If year and month are present and day is missing, set day to the last day of month.

# **6.7.6 Safety Parameters**

Safety and tolerability endpoints will consist of all adverse events (AEs) reported during the study duration from the date of randomization through Week 12 (End of Study Visit).

Specific AEs are defined below.

Treatment-Emergent Adverse Events (TEAE): Any AE with onset after the first dose of study medication through 56 days after the last dose of study medication.

Serious Adverse Event (SAE): An AE occurring at any dose that results in any of the following outcomes: death, a life-threatening AE, in-patient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect.

Associated with Use of the Study Drug: There is a reasonable possibility that the experience may have been caused by the study drug. If the Investigator does not know whether or not study drug caused the event, then the event will be handled as "related to study drug" for reporting purposes. The determination of whether an AE is related to study drug is as follows:

- Related: The AE has a missing, unknown, possible, probable or definite relationship to the study medication.
- Not related: The AE is unlikely or definitely unrelated to the study drug.

# 6.7.7 Missing Start and Stop Dates for Adverse Events

#### Start date:

o If start date is completely missing, start date is set to date of first dose.





Version 1

### Protocol: RB244-001 STATISTICAL ANALYSIS PLAN


Office of the confidential of th

present, and month is missing):

If year = year of first dose, then set month and day to month and day of first dose.

If year < year of first dose, then set month and day to December 31st.

If year > year of first dose, then set month and day to January 1st.

o If month and year are present and day is missing:

If year = year of first dose and

- If month = month of first dose, then set day to day of first dose date
- If month < month of first dose, then set day to last day of month.
- If month > month of first dose, then set day to 1st day of month.

If year < year of first dose, then set day to last day of month.

If year > year of first dose, then set day to 1st day of month.

# Stop date:

If the outcome of the AE was ongoing or unknown, then the rules outlined below will not be applied.

- o If stop date is completely missing, stop date is set to date of study discontinuation.
- o If (year is present, and month and day are missing) or (year and day are present, and month is missing):

If year = year of study discontinuation, then set month and day to month and day of study discontinuation.

If year < year of study discontinuation, then set month and day to December 31st.

If year > year of study discontinuation, then set month and day to December 31st.

o If month and year are present and day is missing:

If year = year of study discontinuation and

- If month = month of study discontinuation, then set day to day of study discontinuation date.
- If month < month of study discontinuation, then set day to last day of month.
- If month > month of study discontinuation, then set day to last day of month.

If year < year of study discontinuation, then set day to last day of month. If year > year of study discontinuation, then set day to last day of month.





# 7 DATA ANALYSES

The data analysis will be conducted on all participant data when the trial ends. Subjects will be pooled across all sites. Data will be presented by treatment group and overall. Categorical variables will be summarized by frequency distributions (number and percentages of subjects) and continuous variables will be summarized by descriptive statistics (mean, standard deviation, etc.).

Adverse events will be summarized by treatment group using the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment-emergent AEs (TEAEs), treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, discontinuations due to AEs, and AEs Grade 3 severity. By-subject listings will be provided for any deaths, SAEs, and AEs leading to discontinuation.

Descriptive statistics for each treatment group will be provided for clinical laboratory values (e.g., hematology, serum chemistry, and urinalysis) and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation. Abnormal clinical laboratory values will be listed.

All data will be provided in by-subject listings.

# 7.1 Subjects Disposition

The subject disposition summary will include the number screened, the number of screen failures, the number enrolled, the number in each patient population for analysis, the number who completed the study, the number who discontinued the study and reason for discontinuation from the study. Disposition data will be summarized by treatment and overall.

A by-subject data listing of study completion information including the reason for study discontinuation will be presented. A by-subject listing of inclusion/exclusion criteria not met will also be presented.

### 7.2 Protocol Deviations

A summary of all protocol deviations on ITT population by type will be generated. Protocol deviation data will be summarized by treatment and overall. A by-subject data listing of protocol deviations will also be presented.

All protocol deviations will be presented in a data listing.





# 7.3 Demographic and Baseline Characteristics

Demographic and baseline characteristic data summarization will be performed to descriptively assess the comparability of treatment groups. Data to be tabulated will include age, race, ethnicity, height, weight, and BMI, as well as baseline characteristics related to medical history, including hypertension, diabetes, smoking history.

# 7.4 Study Drug Exposure

At Baseline visit, Subjects will receive a kit containing (2) two 30 ml white bottles. Each bottle will be used for 2 weeks. At Week 4, subjects will return the used bottles from the kit and will be issued a new kit of two 30mL white bottles to be used from Week 4 through Week 8.

The cumulative amount of study drug exposure will be estimated by calculating the difference between the weight of the 2 bottles of drug at the time the drug was dispensed at Baseline/Week 4 and the weight of the 2 bottles at Week 4/Week 8. Differences will be summed together.

The amount of product used per day will be estimated by dividing the change by the number of days the subject was on treatment. These weights will be compared to the weight of the product that would be used if the subject was compliant with the protocol. Percent compliance will be calculated as follows:



The number of days the subject administered study drug, the amount of product used, and the percent compliance will be summarized by treatment group and presented in a by-subject data listing. The subject listing will also include by-visit IP weights. Percent compliance will be calculated only for subjects who returned the study drug at the end of the treatment. In the listing, subjects who withdrew from the study early will be flagged.

# 7.5 Medical History

A by subject data listing of medical history will be presented. Medical history will be coded using MedDRA v20.0, and the number and percentage of patients experiencing at least 1 such diagnosis by MedDRA System Organ Class (SOC) and preferred term (PT) will be reported.





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN


## 7.6 Concomitant Medication

Concomitant medications will be coded using the World Health Organization (WHO) dictionary. Results will be tabulated by anatomic therapeutic class (ATC) and preferred term.

This data will be summarized by treatment group. Previous and concomitant medications will be presented in a data listing.

# 7.7 Vital Signs and Physical Examination

Vital sign measurements will be presented for each subject in a data listing. Systolic blood pressure, diastolic blood pressure, heart rate, and weight will be summarized as actual value and change from baseline by visit.

All physical examination findings will be presented in a data listing.

# 7.8 Laboratory Data

Clinical laboratory values will be expressed in SI units reported by the central laboratory.

The actual value and change from screening will be summarized for each clinical chemistry, hematology, lipid panel, HbA1C and urinalysis parameters and by each visit. In the event of repeat values, the last non-missing value per visit will be used.

Sample for Serology was collected only at Baseline. Hence Serology data will be only provided in a listing.

All laboratory data will be also provided in data listings. Values outside of the lab parameter's normal range will be flagged as high, low, or abnormal based on the range of the test.

### 7.9 Visit Windows

It is expected that all visits should occur according to the protocol schedule. All data will be tabulated per the evaluation visit as recorded on the CRF even if the assessment is outside of the visit window. In data listings, the relative day of all dates will be presented.

# 8 STATISTICAL ANALYSES

# 8.1 Sample Size Determination

Sample size of 104 randomized 1:1 Active to Vehicle based on 80% power to detect 33% IGA response in Active group versus 10% in the Vehicle group, with two-sided test and alpha =0.05. Until mentioned all alpha value is set at 0.05.





Version 1

14-Feb-19

Protocol: RB244-001 STATISTICAL ANALYSIS PLAN

# 8.2 Safety Analysis

CLINICAL RESEARCH OPTIMIZED™

Safety analyses will be conducted using the Safety population

# 8.2.1 Primary Safety Endpoint

Assess the safety and tolerability of B244 applied twice daily to the face for 8 weeks in subjects with mild to moderate rosacea.

The reporting of safety data is descriptive and will include all subjects who receive at least one dose of investigational product. The variables for safety endpoints are number of subjects with AEs, SAEs, vital signs measurements, clinical chemistry and hematology. AEs will be summarized based on the frequency of AEs and their severity for all treated subjects. All AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA) and summarized by treatment group. Data will be summarized using preferred term and primary system organ class.

If a subject experiences multiple events that map to a single preferred term, the greatest severity and strongest Investigator assessment of relation to investigational product will be assigned to the preferred term for the appropriate summaries. Should an event have a missing severity or relationship, it will be classified as having the highest severity and/or strongest relationship to investigational product.

Summaries of AEs will include any AEs reported beginning with the first dose of investigational product on Day 1. The occurrence of adverse events will be summarized by treatment group using preferred terms, system organ classifications, and severity. Separate summaries of serious adverse events, adverse events related to investigational product, and events leading to the discontinuation of investigational product will be generated. All adverse events reported will be listed for individual subjects showing both verbatim and preferred terms.

# 8.3 Efficacy Analysis

All efficacy endpoints are exploratory endpoints.

Assessment of Superiority:

- IGA treatment success, defined as "clear" or "almost clear" with a 2-grade improvement in IGA score from baseline to the end of treatment (Week 8).
- CEA treatment success, defined as "clear" or "almost clear" with a 2-grade improvement in CEA score from baseline to the end of treatment (Week 8).

Superiority will be based on the proportion of subjects for whom treatment was successful. The comparison will be through a continuity-corrected Z-tests. The Evaluable Period for the outcome variables will be weeks 1, 4, 8 and 12. The superiority of the drug over the vehicle will be tested at week 8 based on the probability of





#### Protocol: RB244-001 STATISTICAL ANALYSIS PLAN


> improvement from baseline with a continuity-corrected Z-tests comparing the change from baseline of treatments vs Placebo. For all other evaluable periods, descriptive statistics for the change from baseline will be shown.

> The null and alternative statistical hypotheses for the primary effectiveness endpoints are given by:

> (Ho): The null hypothesis is that the probability of improving (baseline to week 8) with drug T (PrT) is less than or equal to the probability of improving with vehicle (PrV).

```
H o :
       PrT
                -PrPV = VV:
                             PrT
```

(Ha): The alternative hypothesis is that the probability of improving with drug T (PrT) is greater than to the probability of improving with vehicle (PrV).

```
Ha: PrT > PrV; PrT - PrV = 0
```

For testing the superiority, the following SAS code will be used:

```
proc freq data = dataset;
tables treat*outcome/riskdiff (equal);
run;
```

Change of Skindex 16 patient reported outcome from Baseline to Week 1, Week 4, Week 8 and Week 12

The change from baseline score of Skindex-16 will be compared among treatments at Week 12 using an ANOVA, to test the Skindex 16 score change from Baseline to Week 12 for the two treatments. Also, descriptive stats will be used to assess the change from Baseline to Week 1, 4, 8 & 12.

- Change of IGA score at Baseline to Week 1, Week 4, Week 8 and Week 12.
- Change of CEA score at Baseline to Week 1, Week 4, Week 8 and Week 12.
- Change of PSA score at Baseline to Week 1, Week 4, Week 8 and Week 12.

Descriptive stats will be used to show the change from Baseline to Week 1, 4, 8 & 12.

#### **Sensitivity Analysis** 8.4

A sensitivity analysis will be performed by Multiple Imputation Regression Analysis using the following factors: treatment, age, gender, race, baseline IGA, baseline CEA, baseline PSA, smokers/non-smokers and the results of the same variable from previous visits. The Proc MI SAS code will be used to perform the analysis based on the mentioned factors.






# 9 REFERENCES

- Protocol Number: RB244-001, VER 4.0 "A Vehicle-Controlled, Double-Blind, Randomized Phase II Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects with Mild to Moderate Rosacea."
- Wang, Wei. (1988, October 28). Calculating Age in One Line of Code. Paper presented at annual meeting of Northeast SAS Users Group, New York, New York. Paper retrieved from <a href="http://www.lexjansen.com/nesug/nesug01/cc/cc4022.pdf">http://www.lexjansen.com/nesug/nesug01/cc/cc4022.pdf</a>.
- DE MARS, A. (2018). "Mixed Reviews": An Introduction to Proc Mixed. Retrieved from <a href="http://www.hawaii.edu/hisug/pdf/AnnMariaprocmixed.pdf">http://www.hawaii.edu/hisug/pdf/AnnMariaprocmixed.pdf</a>
- Moser, E. (2018). Repeated Measures Modeling with PROC MIXED. Retrieved from http://www2.sas.com/proceedings/sugi29/188-29.pdf





### **10 APPENDIX**

### 10.1 APPENDIX A: Tables

### **10.1.1 General**

| Display Number | Title | Population | Unique/Repeat |
|---|---|---|---|
| 14.1.1.1 | Subject Enrollment and Disposition | All Subjects | Unique |
| 14.1.1.2 | Subject Enrollment and Disposition | Enrolled Subjects | Repeat |
| 14.1.1.3 | Analysis Population and Exclusions | All Subjects | Unique |
| 14.1.2.1 | Summary of Protocol Deviations (PD)/Violations (PV) | mITT | Unique |
| 14.1.2.2 | Summary of Protocol Deviations (PD)/Violations (PV) | Safety | Repeat |
| 14.1.3.1 | Summary of Demographic and Baseline<br>Characteristics | mITT | Unique |
| 14.1.3.2 | Summary of Demographic and Baseline<br>Characteristics | PP | Repeat |
| 14.1.3.3 | Summary of Demographic and Baseline<br>Characteristics | Safety | Repeat |
| 14.1.4.1 | Summary of Vital Sign | mITT | Unique |
| 14.1.4.2 | Summary of Vital Sign | PP | Repeat |
| 14.1.4.3 | Summary of Vital Sign | Safety | Repeat |
| 14.1.5.1 | Summary of Physical Examination | mITT | Unique |
| 14.1.5.2 | Summary of Physical Examination | PP | Repeat |
| 14.1.5.3 | Summary of Physical Examination | Safety | Repeat |
| 14.1.6 | Summary of Study Drug Accountability: Dose Dispensed & Collected by Visit | Safety | Unique |
| 14.1.7.1 | Summary of Study Drug Compliance | Safety | Unique |
| 14.1.7.2 | Summary of Percent Compliance based on<br>Cumulative Net Weight of Study Drug | Safety | Unique |
| 14.1.8 | Summary of Prior Medications | Safety | Unique |
| 14.1.9 | Summary of Concomitant Medications | Safety | Unique |
| 14.1.10 | Summary of Medical History | Safety | Unique |
| 14.1.11 | Summary of Substance Abuse | Safety | Unique |
| 14.1.12 | Summary of Dairy Details | Safety | Unique |






#### STATISTICAL ANALYSIS PLAN


Table 14.1.1.1 Subject Enrollment and Disposition

## All Subjects

| Disposition | B244 Topical Spray<br>n (%) | Placebo<br>n (%) | All Patients<br>n (%) |
|---|---|---|---|
| Screened | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Randomized | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treated | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed Study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed Week 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed Week 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed Week 8 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed Week 12 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Screen Failure | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal of consent | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| In the opinion of the Investigator, it is not in<br>the subject's best interests to continue in the<br>study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Occurrence of an Adverse Event (AE) or<br>Serious Adverse Event (SAE), which, in the<br>opinion of the Investigator warrants<br>discontinuation of the subject from the study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Significant non-compliance with study procedures that would interfere with the study results or increase the subject's risks in the study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject is deemed to be a treatment failure, which is defined as worsening of condition and requiring alternate or supplemental therapy | xx (xx.x) | xx (xx.x) | xx (xx.x) |





| Protocol: RB244-001<br>Confidential | STATISTICA | L ANALYSIS PLAN | | Version 1<br>14-Feb-19 |
|---|---|---|---|---|
| for the treatment of external during the study | anogenital warts | | | |
| The subject's medication cod | e is unblinded | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject did not meet, or no lo entry criteria | onger meets, the | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| The subject is lost to follow-u | р | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Investigator discretion | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NOTE: The percentages are b | agad on the | | Spanish at Data | DD MMM VVVV |

NOTE: The percentages are based on the number of randomized subjects.

Snapshot Data DD-MMM-YYYY

Program Name: <Pgm name> Source: <Dataset>

Repeat as 14.1.1.2 for Enrolled Subject.

Table 14.1.1.3 Analysis Population and Exclusions All Subjects

| Number of Subjects | B244 Topical Spray n (%) | Placebo<br>n (%) | All Patients n (%) |
|---|---|---|---|
| Enrolled | XX | XX | XX |
| Randomized | xx | XX | XX |
| Included in Safety Population | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Reasons for Exclusion from Safety Population | | | |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Included in Full Analysis Set Reasons for Exclusion from Safety Population | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Reasons for Exclusion from Safety Population | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |





| Protocol: RB244-001<br>Confidential | STATISTICAL ANALYSIS PLAN | | Version 1<br>14-Feb-19 |
|---|---|---|---|
| Included in Per Protocol Population Reasons for Exclusion from Per Protocol | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Did not receive randomized therapy | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |

NOTE: The percentages are based on the number of randomized subjects.

Snapshot Data DD-MMM-YYYY

Program Name: <Pgm name>

C .....

Source: <Dataset>

Table 14.1.2.1 Summary of Protocol Deviations (PD)/Violations (PV) mITT Population

| | | | | All |
|---------------------|---------|--------------------|---------|----------|
| | | B244 Topical Spray | Placebo | Patients |
| Deviation/Violation | PD/PV | n (%) | n (%) | n (%) |
| Description of | "PD" or | n (%) | n (%) | n (%) |
| Violation/deviation | "PV" | XX | XX | XX |

N: Number of Patients

Xx: Number of deviations/violations

Source: <Dataset> Snapshot Data DD-MMM-YYYY

Program Name: <Pgm name>

Repeat for Safety Population

### Table 14.1.3.1 Summary of Demographic and Baseline Characteristics mITT Population

| | | B244 Topical Spray | Placebo | All Patients |
|----------|-----------|--------------------|--------------|--------------|
| Variable | Statistic | n (%) | n (%) | n (%) |
| Age | N | XX | XX | XX |
| | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | xx.x(xx.xxx) |







| Protocol: RB244-001 STATISTICAL ANALYSIS PLAN Confidential | | | | Version 1<br>14-Feb-19 |
|---|---|---|---|---|
| Confidential | | B244 Topical Spray | Placebo | All Patients |
| Variable | Statistic | n (%) | n (%) | n (%) |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Sex | | | | |
| Male | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Female | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Ethnicity | , , | , , | | |
| Hispanic or Latino | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Not Hispanic or Latino | N (%) | xx(xx.x) | xx (xx.x) | xx(xx.x) |
| Race | | | | |
| American Indian or | | | | |
| Alaskan Native | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Asian | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Black or African | , , | , , | ` , | ` ′ |
| American | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Native Hawaiian or | , , | , , | ` , | ` ′ |
| Other Pacific Islander | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| White | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Other | N (%) | xx(xx.x) | xx (xx.x) | xx (xx.x) |

Snapshot Data DD-MMM-YYYY Program Name: <Pgm name>

Source: <Dataset>

Repeat for PP and Safety population

Table 14.1.4.1 Summary of Vital Signs, mITT Population

| Visit | Vital Sign | Statistic | B244 Topical<br>Spray<br>n (%) | Placebo<br>n (%) | All Patients n (%) |
|---|---|---|---|---|---|
| Baseline | Height | N | XX | XX | XX |
| | | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | XX.X |
| | | | | | (xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Weight | N | XX | XX | XX |
| | | | | | XX.X |
| | | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | (xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Temperature | N | XX | XX | XX |






#### STATISTICAL ANALYSIS PLAN


| uciitiai | | | | | 14-1-60-1 |
|---|---|---|---|---|---|
| | | | B244 Topical | | |
| | | | Spray | Placebo | All Patients |
| Visit | Vital Sign | Statistic | n (%) | n (%) | n (%) |
| | | | | | XX.X |
| | | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | (xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Heart Rate | N | XX | XX | XX |
| | | | | | XX.X |
| | | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | (xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Systolic BP | N | XX | XX | XX |
| | | | | | XX.X |
| | | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | (xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Diastolic BP | N | XX | XX | XX |
| | | | | | XX.X |
| | | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | (xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Repeat for | | | | | |
| every visit | | | | | |
| showing | | | | | |
| Change from | | | | | |
| Baseline | | | | | |

Snapshot Data DD-MMM-YYYY

Repeat for PP and Safety population

### Table 14.1.5.1 Summary of Physical Examination, mITT Population

| | | | B244 Topical | | |
|---|---|---|---|---|---|
| | | | Spray | Placebo | All Patients |
| Visit | Physical Examination | Statistic | n (%) | n (%) | n (%) |
| Baseline | Height | N | XX | XX | XX |






#### STATISTICAL ANALYSIS PLAN


| Communication | | | | | 1110017 |
|---|---|---|---|---|---|
| | | | B244 Topical | | |
| | | | Spray | Placebo | All Patients |
| Visit | Physical Examination | Statistic | n (%) | n (%) | n (%) |
| | | Mean (SD) | xx.x (xx.xxx) | XX.X | xx.x (xx.xxx) |
| | | | | (xx.xxx) | |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Weight | N | XX | XX | XX |
| | | | | XX.X | |
| | | Mean (SD) | xx.x (xx.xxx) | (xx.xxx) | xx.x (xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | General Appearance | | | | |
| | Normal | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Abnormal | N (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| | Heart Cardiovascular | | | | |
| | Normal | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Abnormal | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Lungs | | | | |
| | Normal | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Abnormal | N (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| | Gastrointestinal | | | | |
| | Normal | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Abnormal | N (%) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| | Ear/Nose/Throat | | | | |
| | Normal | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Abnormal | N (%) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| | Extremities | | | | |
| | Normal | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Abnormal | N (%) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| | Skin | | | | |
| | Normal | N (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| | Abnormal | N (%) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Repeat for | | | | | |
| every week | | | | | |

CRF pages 05-06 Source: <Dataset> Snapshot Data DD-MMM-YYYY
Program Name: <Pgm name>

Repeat for PP and Safety populations






### Table 14.1.6 Summary of Study Drug Accountability: Dose Dispensed & Collected by Visit Safety Population

| | | B244 Topical Spray | Placebo | All Patients |
|---|---|---|---|---|
| Weight of the Dose | Statistic | n (%) | n (%) | n (%) |
| Dose Dispensed | N | XX | XX | XX |
| | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | xx.x(xx.xxx) |
| | CV | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Repeat for Dose Collected | | | | |
| Total Dose Dispensed | N | XX | XX | XX |
| - | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | xx.x(xx.xxx) |
| | CV | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Repeat for Total Dose Collected | | | | |

N: Number of Patients CRF pages 28-30 Snapshot Data DD-MMM-YYYY Source: <Dataset> Program Name: <Pgm name>

Table 14.1.7.1 Summary of Study Drug Compliance Safety Population

| 5. | arety reparation | | |
|---|---|---|---|
| | B244 Topical | | All |
| | Spray | Placebo | Patients |
| Statistic | n (%) | n (%) | n (%) |
| h | | | |
| N (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| N (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| N | xx | XX | XX |
| Mean (SD) | xx.x (xx.xxx) | xx.x (xx.xxx) | xx.x<br>(xx.xxx) |
| CV | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| | Statistic h N (%) N (%) N (%) CV | B244 Topical Spray n (%) | Statistic Spray n (%) Placebo n (%) h N (%) xx (xx.x) xx (xx.x) N (%) xx (xx.x) xx (xx.x) N (%) xx (xx.x) xx (xx.xx) N (%) xx (xx.xx) xx (xx.xx) CV xx.x (xx.xxx) xx.x |







| Protocol: RB244-001<br>Confidential | STATISTICAL ANALYSIS PLAN | | | | Version 1<br>14-Feb-19 |
|---|---|---|---|---|---|
| | Min, Max | XX.X, XX.X | XX.X | X, XX.X | XX.X, |
| | | | | | XX.X |
| Applications: Number of | of applications per pa | atients/day | | Snapshot Dat | ta DD-MMM- |
| (expected 4 Pumps twi | ce a Day) | | | • | YYYY |
| | | ( | CRF pages 30 | | |
| Compliance: The expec | ted amount of study | drug used | | Program | Name: <pgm< td=""></pgm<> |
| per week is approximat | ely 7.84 g/week for | 8 | Source: | | name> |
| sprays/application per | day | < | <dataset></dataset> | | |

Table 14.1.7.2
Summary of Percent Compliance based on Cumulative Net Weight of Study Drug
Safety Population
B244 Topical

| | | D2 <del>44</del> 10picai | | |
|---|---|---|---|---|
| | | Spray | Placebo | All Patients |
| | Statistic | n (%) | n (%) | n (%) |
| Cumulative Net Weight of Study Drug | | | | |
| , , | N | XX | XX | XX |
| | Mean (SD) | xx.x(xx.xxx) | xx.x (xx.xxx) | xx.x (xx.xxx) |
| | CV | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Percent Compliance greater than 50% | | | | |
| Yes | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| No | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

Applications: Number of applications per patients/day (expected 4 Pumps twice a Day)

Snapshot Data DD-MMM-YYYY

The cumulative amount of study drug exposure

will be estimated by calculating the difference between the weight of the 2 bottles of drug at the time the drug was dispensed at Baseline/Week 4 and the weight of the 2 bottles at Week 4/Week 8. Differences will be summed together.

Program Name: <Pgm name>

Source: <Dataset>

CRF pages 30

% Compliance: The net weight of study drug divided by 1.12g /Day \* Number of Days in the Study





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN

Version 1 14-Feb-19 Confidential

Table 14.1.8 Summary of Prior Medications, Safety Population

| WHO-DD ATC Class Level 1<br>WHO-DD ATC Class Level 2 | B244 Topical<br>Spray | Placebo | All Patients |
|---|---|---|---|
| WHO-DD Preferred Term | n (%) | n (%) | n (%) |
| Number of subjects with at least one prior medication | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| WHO-DD ATC Class Level 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| WHO-DD ATC Class Level 2 | xx(xx.x) | xx (xx.x) | xx(xx.x) |
| WHO-DD Preferred Term 1 | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| WHO-DD Preferred Term 2 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| etc. | | | |
| WHO-DD ATC Class Level 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| WHO-DD ATC Class Level 2 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD Preferred Term 1 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD Preferred Term 2 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| etc. | | | |

NOTE: The percentages are based on the

Snapshot Data DD-MMM-YYYY

number of Safety Population.

CRF page 11

Program Name: <Pgm name> Source: <Dataset>

Table 14.1.9 Summary of Concomitant Medications, Safety Population

| WHO-DD ATC Class Level 1 | B244 Topical | | All |
|---|---|---|---|
| WHO-DD ATC Class Level 2 | Spray | Placebo | Patients |
| WHO-DD Preferred Term | n (%) | n (%) | n (%) |
| Number of subjects with at least one concomitant medication | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD ATC Class Level 1 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD ATC Class Level 2 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD Preferred Term 1 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD Preferred Term 2 | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| etc. | | | |
| WHO-DD ATC Class Level 1 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD ATC Class Level 2 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD Preferred Term 1 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD Preferred Term 2 | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| etc. | | | |






NOTE: The percentages are based on the

Snapshot Data DD-MMM-YYYY

number of Safety Population.

CRF pages 12-13

Source: <Dataset>

Program Name: <Pgm name>

### Table 14.1.10 Summary of Medical History Safety Population

| WHO-DD SOC | B244 Topical<br>Spray | Placebo | All Patients |
|---|---|---|---|
| WHO-DD Preferred Term | n (%) | n (%) | n (%) |
| Number of subjects with at least one Medical History | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| WHO-DD SOC | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| WHO-DD Preferred Term | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| WHO-DD Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| WHO-DD Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| etc. | | | |

NOTE: The percentages are based on the number of Safety Population.

Snapshot Data DD-MMM-YYYY

CRF pages

Source: <Dataset>

Program Name: <Pgm name>

### Table 14.1.11 Summary of Substance Abuse Safety Population

| | Statistics | B244<br>Topical<br>Spray<br>N (xxx) | Placebo<br>N (xxx) | All Patients<br>N (xxx) |
|---|---|---|---|---|
| Total Number of Substance Abuse | n | XX<br>XX | XX<br>XX | XX<br>XX |
| | | XX | XX | XX |
| Number of Subjects with Substance<br>Abuse History | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | xx (xx.x) | xx (xx.x) | xx (xx.x) |





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN Version 1 Confidential 14-Feb-19

> xx(xx.x)xx(xx.x)xx(xx.x)

NOTE: The percentages are based on the

Snapshot Data DD-MMM-YYYY

number of Safety Population.

CRF pages Source: <Dataset>

Program Name: <Pgm name>

Table 14.1.12 Summary of Diary Details Safety Population

| | Statistics | B244 Topical<br>Spray<br>N (xxx) | Placebo<br>N (xxx) | All Patients<br>N (xxx) |
|---|---|---|---|---|
| Number of Subjects with diary Dispensed | n | XX | XX | XX |
| Number of Subjects with diary Collected | n | XX | XX | XX |
| | | XX | XX | XX |
| Number of Subjects with Sunscreen use | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Subjects with Makeup use | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

NOTE: The percentages are based on the number of Safety Population.

Snapshot Data DD-MMM-YYYY

CRF pages

Source: <Dataset> Program Name: <Pgm name>






### 10.1.2 Efficacy

| Display Number | Title | Population | Unique/Repeat |
|---|---|---|---|
| 14.2.1.1 | Change from baseline in IGA score by Visit | mITT | Unique |
| 14.2.1.2 | Change from baseline in IGA score by Visit | PP | Repeat |
| 14.2.2.1 | Change from baseline in CEA score by Visit | mITT | Repeat |
| 14.2.2.2 | Change from baseline in CEA score by Visit | PP | Repeat |
| 14.2.3.1 | Change from baseline in PSA score by Visit | mITT | Repeat |
| 14.2.3.2 | Change from baseline in PSA score by Visit | PP | Repeat |
| 14.2.4.1 | Summary of Change from baseline in Skindex 16 score by Visit | mITT | Unique |
| 14.2.4.2 | Summary of Change from baseline in Skindex 16 score by Visit | PP | Repeat |
| 14.2.5 | Summary of Sensitivity Analysis | mITT | Unique |
| 14.2.6.1 | Summary of 2-grade improvement in IGA score from baseline to the end of treatment (Week 8). | mITT | Unique |
| 14.2.6.2 | Summary of 2-grade improvement in IGA score from baseline to the end of treatment (Week 8). | PP | Repeat |
| 14.2.7.1 | Summary of 2-grade improvement in CEA score from baseline to the end of treatment (Week 8). | mITT | Repeat |
| 14.2.7.2 | Summary of 2-grade improvement in CEA score from baseline to the end of treatment (Week 8). | PP | Repeat |
| 14.2.8.1 | Summary of Treatment success with IGA score of 0/1 from Baseline to End of Treatment. | mITT | Unique |
| 14.2.8.2 | Summary of Treatment success with IGA score of 0/1 from Baseline to End of Treatment. | PP | Repeat |
| 14.2.9.1 | Summary of Treatment success with CEA score of 0/1 from Baseline to End of Treatment. | mITT | Repeat |
| 14.2.9.2 | Summary of Treatment success with CEA score of 0/1 from Baseline to End of Treatment. | PP | Repeat |






### Table 14.2.1.1 Change from baseline in IGA Score by Visit. mITT Population

| | B244 Topical | | |
|---------------------------|--------------|---------|--------------|
| | Spray | Placebo | All Patients |
| Visit | N (xxx) | N (xxx) | N (xxx) |
| W71- 1 | | | |
| Week 1 | | | |
| Change from Baseline | | | |
| 1-grade | n (%) | | |
| 2-grade | n (%) | | |
| 3-grade | n (%) | | |
| Repeat for all the visits | | | |

CRF pages
Source: <Dataset>

Snapshot Data DD-MMM-YYYY

Program Name: <Pgm name>

Repeat for CEA and PSA for mITT & PP population.

Table 14.2.4.1 Summary of Change from baseline in Skindex 16 score by Visit mITT Population

| | B244 Topical<br>Spray | Placebo | All Patients |
|---|---|---|---|
| Visit | N (xxx) | N (xxx) | N (xxx) |
| Baseline | | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x (xx.xxx) | xx.x(xx.xxx) | xx.x(xx.xxx) |
| CV | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Change from Baseline at Week 1 | | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | xx.x(xx.xxx) |
| CV | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Repeat for All weeks | | | |
| Final Analysis for Week 12 | | | |
| Differences of LS Means | | | X.XXXX |





SE x.xxxx

CI P-value (x.xxxx, x.xxxx)

SE: Standard Error of the LS Means

P- Value: Probability of Change from Baseline at Week 12

CRF pages Snapshot Data DD-MMM-YYYY

Source: <Dataset> Program Name: <Pgm name>

Repeat for PP population.

# Table 14.2.5 Summary of Sensitivity Analysis for the Absolute Scores of IGA, CEA & PSA mITT Population

| | B244 Topical<br>Spray | Placebo | All Patients |
|---|---|---|---|
| Imputation | N (xxx) | N (xxx) | N (xxx) |
| Imputation#1 | | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x(xx.xxx) | xx.x (xx.xxx) | xx.x (xx.xxx) |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Imputation#2 | | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | xx.x(xx.xxx) |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Repeat for all imputations | | | |
| Analysis Summary | | | |
| Parameter1 | | | xx.x (xx.xxx) |
| Mean (SD) | | | X.XX, X.XX |
| CI | | | X.XXX |
| P-Value | | | |
| Parameter2 | | | |
| Parameter3 | | | |

SD: Standard Error of the Parameters

P- Value: Significance of the Parameters effecting the imputation

CRF pages
Source: <Dataset>

Snapshot Data DD-MMM-YYYY
Program Name: <Pgm name>






#### STATISTICAL ANALYSIS PLAN


Table 14.2.6.1
Summary of 2-grade improvement in IGA score from baseline to the end of treatment (Week 8).
mITT Population

| | B244 Topical<br>Spray<br>N (xxx) | Placebo<br>N (xxx) | All Patients<br>N (xxx) |
|---|---|---|---|
| Subjects with 2-Grade improvement from Baseline to Week 8 | n (%) | n (%) | n (%) |
| Risk Difference<br>CI<br>One Sided P-value | | | X.XXX<br>(X.XX, X.XX)<br>X.XXXX |

CI: Confidence Interval

P-value: Probability of Superiority from the Placebo

Snapshot Data DD-MMM-YYYY

Program Name: <Pgm name>

Repeat for PP Population and for CEA (mITT & PP).

Table 14.2.8.1 Summary of Treatment success with IGA score of 0 or 1. mITT Population

Source: <Dataset>

| | B244 Topical<br>Spray<br>N (xxx) | Placebo<br>N (xxx) | All Patients<br>N (xxx) |
|---|---|---|---|
| Subjects with IGA Score of 0/1 at End of Treatment | n (%) | n (%) | n (%) |
| CI<br>P-value | | | (x.xx, x.xx)<br>x.xxxx |

CI: Confidence Interval

P-value: Probability of achieving Treatment Success defined as a score of 0/1.

Snapshot Data DD-MMM-YYYY

Source: <Dataset> Program Name: <Pgm name>

Repeat for PP Population and for CEA (mITT & PP)






### **10.1.3** Safety

| Display Number | Title | Population | Unique/Repeat |
|---|---|---|---|
| 14.3.1 | Overall Summary of Treatment Emergent | Safety | Unique |
| | Adverse Events | | |
| 14.3.1.1 | Summary of Treatment Emergent Adverse | Safety | Unique |
| | Events by System Organ Class and | | |
| | Preferred Term | | |
| 14.3.1.2 | Summary of Treatment Emergent Adverse | Safety | Repeat |
| | Events by System Organ Class, Preferred | | |
| | Term and Severity | | |
| 14.3.1.3 | Summary of Treatment Emergent Adverse | Safety | Repeat |
| | Events by System Organ Class, Preferred | | |
| | Term and Relationship to Study Drug | | |
| 14.3.2 | Summary of Serious Adverse Events by | Safety | Repeat |
| | System Organ Class and Preferred Term | - | |
| 14.3.3 | Summary of Deaths | Safety | Unique |

Table 14.3.1 Overall Summary of Treatment Emergent Adverse Events. Safety Population

| | Statistics | B244 Topical<br>Spray<br>n (%) | Placebo<br>n (%) | All Patients n (%) |
|---|---|---|---|---|
| T-4-1 Nh | NI | | | |
| Total Number of TEAEs | N | XX | XX | XX |
| Total Number of TESAEs | N | XX | XX | XX |
| Number of Subjects with: At Least One TEAE At Least One Related TEAE At Least One Severe (Grade 3) TEAE At Least One TEAE Leading to Discontinuation At Least One TEAE Leading to Death At Least One TESAE At Least One Related TESAE | n (%) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

CRF pages Source: <Dataset> Snapshot Data DD-MMM-YYYY
Program Name: <Pgm name>






#### STATISTICAL ANALYSIS PLAN


Table 14.3.1.1

### Overall Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

| | Statistics | B244 Topical<br>Spray<br>n (%) | Placebo<br>n (%) | All Patients<br>n (%) |
|---|---|---|---|---|
| Total Number of TEAEs | n | xx | xx | XX |
| Number of Subjects with at Least One TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #1 Preferred Term #1 Preferred Term #2 Preferred Term #3 etc. | n (%)<br>n (%)<br>n (%)<br>n (%) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| System Organ Class #2 Preferred Term #1 Preferred Term #2 Preferred Term #3 etc. | n (%)<br>n (%)<br>n (%)<br>n (%) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

CRF pages Source: <Dataset> Snapshot Data DD-MMM-YYYY Program Name: <Pgm name>

Table 14.3.1.2

# Overall Summary of Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Severity **Safety Population** B244 Topical

| | | | D277 Topical | | |
|---|---|---|---|---|---|
| | | | Spray | Placebo | All Patients |
| | Statistics | Severity | N (xxx) | N (xxx) | N (xxx) |
| Total Number of TEAEs | n | Mild | XX | XX | XX |
| | | Moderate | XX | XX | XX |
| | | Severe | XX | XX | XX |
| | | Total | XX | XX | XX |
| Number of Subjects with at Least One TEAE | n (%) | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| · | , , | Moderate | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| | | Severe | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| | | Total | xx(xx.x) | xx (xx.x) | xx(xx.x) |





Snapshot Data DD-MMM-YYYY Program Name: <Pgm name>

| Protocol: RB244-001<br>Confidential | STATISTICAL ANALYSIS PLAN | | | Version 1<br>14-Feb-19 | |
|---|---|---|---|---|---|
| System Organ Class #1 | n (%) | Mild<br>Moderate<br>Severe<br>Total | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Preferred Term #1 | n (%) | Mild<br>Moderate<br>Severe<br>Total | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| etc. | | | () | () | () |

CRF pages

Source: <Dataset>

Table 14.3.1.3 Overall Summary of Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Relationship to Study Drug Safety Population

| | Statistics | Relationship | B244<br>Topical<br>Spray<br>N (xxx) | Placebo<br>N (xxx) | All Patients<br>N (xxx) |
|---|---|---|---|---|---|
| Total Number of TEAEs | n | Not Related | XX | xx | XX |
| | | Related | XX | XX | XX |
| | | Total | XX | XX | XX |
| Number of Subjects with at Least One TEAE | n (%) | Not Related | xx (xx.x) | xx (xx.x) | ) xx (xx.x) |
| · | . , | Related | xx (xx.x) | xx (xx.x) | , , |
| | | Total | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| System Organ Class #1 | n (%) | Not Related | xx (xx.x) | xx (xx.x) | ) xx (xx.x) |
| , . | , , | Related | xx (xx.x) | xx (xx.x) | , , |
| | | Total | xx (xx.x) | xx (xx.x) | ` ′ |
| Preferred Term #1 | n (%) | Not Related | xx (xx.x) | xx (xx.x) | ) xx (xx.x) |
| Troining Term // 1 | 11 (70) | Related | XX (XX.X) $XX (XX.X)$ | XX (XX.X) | ` / |
| | | Total | XX (XX.X) | XX (XX.X) | ` / |
| etc. | | 10111 | AA (AA.A) | AA (AA.A) | , AA (AA.A) |

CRF pages Source: <Dataset> Snapshot Data DD-MMM-YYYY Program Name: <Pgm name>






#### STATISTICAL ANALYSIS PLAN


Table 14.3.2 Summary of Serious Adverse Events by System Organ Class and Preferred Term Safety Population

| | Statistics | Relationship | B244 Topical<br>Spray<br>N (xxx) | Placebo<br>N (xxx) | All<br>Patients<br>N (xxx) |
|---|---|---|---|---|---|
| Total Number of SAEs | n | Yes | XX | XX | XX |
| | | No | XX | XX | XX |
| | | Total | XX | XX | XX |
| Number of Subjects with at Least One SAE | n (%) | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | ( ) | No | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| | | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #1 | n (%) | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| , , | . , | No | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| | | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #1 | n (%) | Yes | vv (vv v) | vv (vv v) | vv (vv v) |
| Freieneu reim#1 | 11 (70) | No | xx (xx.x)<br>xx (xx.x) | XX (XX.X) | XX (XX.X) |
| | | Total | xx(xx.x)<br>xx(xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| etc. | | | | | |
| | CRF pages | | Snapshot Data DD-l | $MMM-YYY\overline{Y}$ | |

CRF pages Source: <Dataset> Snapshot Data DD-MMM-YYYY
Program Name: <Pgm name>

Table 14.3.3 Summary of Deaths Safety Population

| | | B244 Topical | | |
|---|---|---|---|---|
| | | Spray | Placebo | All Patients |
| | Statistics | N(xxx) | N (xxx) | N (xxx) |
| Number of deaths | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Related to disease under study | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| AE outcome = death | n (%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Related to disease under study and AE outcome = death | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| and AL outcome – death | | | | |

CRF pages Source: <Dataset> Snapshot Data DD-MMM-YYYY
Program Name: <Pgm name>





Version 1

14-Feb-19

Protocol: RB244-001 STATISTICAL ANALYSIS PLAN

# 10.2 APPENDIX B: Listings

| Display Number | Title | Population |
|---|---|---|
| Listing 16.2.1.1 | Subject Enrollment and Disposition by Study Site | All Subjects |
| Listing 16.2.1.2 | Protocol Deviations (PD)/Violations (PV) | Randomized |
| Listing 16.2.1.3 | Demographic Characteristics | Randomized |
| Listing 16.2.1.4 | Vitals Signs by Subject and Visit | Safety |
| Listing 16.2.1.5 | Physical Examination by Subject | Safety |
| Listing 16.2.1.6 | Drug Exposure and Compliance | Safety |
| Listing 16.2.1.8 | Prior Medications | Safety |
| Listing 16.2.1.9 | Concomitant Medications | Safety |
| Listing 16.2.2.1 | IGA score by Subjects and Visits | Randomized |
| Listing 16.2.2.2 | CEA score by Subjects and Visits | Randomized |
| Listing 16.2.2.3 | PSA score by Subjects and Visits | Randomized |
| Listing 16.2.2.4 | Skindex-16 score by Subjects and Visits | Randomized |
| Listing 16.2.3.1 | Treatment Emergent Adverse Events by System Organ<br>Class, Preferred Term, Severity and Relationship to<br>Study Drug | Safety |
| Listing 16.2.3.2 | Serious Adverse Events by System Organ Class and Preferred Term | Safety |
| Listing 16.2.3.3 | Deaths | Safety |
| Listing 16.2.4.1 | Hematology Parameters | Safety |
| Listing 16.2.4.2 | Clinical Chemistry Parameters | Safety |
| Listing 16.2.4.3 | Urinalysis Parameters | Safety |
| Listing 16.2.4.4 | Serology Parameters | Safety |





Version 1

14-Feb-19

Protocol: RB244-001 STATISTICAL ANALYSIS PLAN

## 10.3 APPENDIX C: Figures

| Display Number | Title | Population |
|---|---|---|
| Figure 14.2.1.1 | Frequency table Change from baseline for IGA score by Visit | mITT |
| Figure 14.2.1.2 | Frequency table Change from baseline for IGA score by Visit | PP |
| Figure 14.2.2.1 | Frequency table Change from baseline for CEA score by Visit | mITT |
| Figure 14.2.2.2 | Frequency table Change from baseline for CEA score by Visit | PP |
| Figure 14.2.3.1 | Frequency table Change from baseline for PSA score by Visit | mITT |
| Figure 14.2.3.2 | Frequency table Change from baseline for PSA score by Visit | PP |
| Figure 14.2.4.1 | Box Plot of Skindex 16 score by Visit | mITT |
| Figure 14.2.4.2 | Box Plot of Skindex 16 score by Visit | PP |
| Figure 14.2.8.1 | Bar Plot for Treatment Success (0/1) for IGA score at Week 12 | mITT |
| Figure 14.2.8.2 | Bar Plot for Treatment Success (0/1) for IGA score at Week 12 | PP |
| Figure 14.2.9.1 | Bar Plot for Treatment Success (0/1) for CEA score at Week 12 | mITT |
| Figure 14.2.9.2 | Bar Plot for Treatment Success (0/1) for CEA score at Week 12 | PP |





STATISTICAL ANALYSIS PLAN Protocol: RB244-001


# STATISTICAL ANALYSIS PLAN PHASE II

**VERSION: 2.0** 

**DATE:** 

**April 02, 2019** 

#### **BASED ON:**

Protocol Version 4.0 Date:07-Jan-19

Data Management Plan Final Version 1.0 Date: 12-Apr-18

### **Study Drug:**

B244 Topical application

#### **Protocol Number:**

RB244-001

### **Study Title:**

Vehicle-Controlled, Double-Blind, Randomized Phase II Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects with Mild to Moderate Rosacea.

### **Sponsor:**

AOBiome, LLC

125 Cambridgepark Drive

Cambridge, MA 02140







Protocol: RB244-001

#### STATISTICAL ANALYSIS PLAN

Version 2


# STATISTICAL ANALYSIS PLAN REVIEW AND APPROVAL

This Statistical Analysis Plan has been prepared in accordance with team reviewers' specifications.

02-Apr-19

| Prepared by: | |
|--------------|-------|
| Mad | . 100 |

Rahul Paul Choudhury, Lead Bio-Statistician

Statistical Review:

Sr. Specialist Bio-Statistician

02 May 2019 Date

Sponsor Review:

Judith Mg-Cashin, M.D, Chief Medical Officer

Spiros Jamas, Sc. D., SVP of Therapeutic Development





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN Version 2 Confidential 02-Apr-19

### PROTOCOL SYNOPSIS

| Study Title | A Vehicle-Controlled, Double-Blind, Randomized Phase II Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects with Mild to Moderate Rosacea. |
|---|---|
| Protocol Number | RB244-001 |
| <b>Development Phase</b> | Phase II |
| Type of Study | Safety Analysis and Superiority of the Study drug over Vehicle |
| Study Medications | <ol> <li>B244 Topical Spray (Test formulation), manufactured by<br/>AOBiome Therapeutics.</li> <li>Vehicle of test product manufactured by AOBiome<br/>Therapeutics.</li> </ol> |
| Name of Active<br>Ingredient | B244 |
| Route of administration | Topical application |
| Sponsor | AOBiome, LLC,125 Cambridgepark Drive, |
| | Cambridge, MA 02140 |
| Study Objectives | PRIMARY |
| | To assess the safety and tolerability of B244 applied twice daily (BID) to the face for 8 weeks in subjects with mild to moderate rosacea. |
| | EXPLORATORY |
| | To assess the efficacy of B244 in subjects with mild to moderate rosacea. |
| | <ul> <li>Proportion of subjects with IGA improvement at Week 8 relative to baseline</li> <li>Proportion of subjects with CEA improvement at Week 8 relative to baseline</li> <li>Change in IGA from Baseline to Week 8</li> <li>Change in CEA from Baseline to Week 8</li> <li>Proportion of Subjects with improvement in IGA or</li> </ul> |





| Protocol: RB244-001<br>Confidential | STATISTICAL ANALYSIS PLAN Version 2 02-Apr-19 |
|---|---|
| | <ul> <li>CEA at Week 1, Week 4, and Week 12.</li> <li>Change in Skindex 16 patient reported outcome from Baseline to Week 1, Week 4, Week 8, and Week 12.</li> <li>Proportion of subjects with change in PSA at Week 1, Week 4, Week 8 and Week 12 from Baseline.</li> <li>Evaluation of Telangiectasia Score at Baseline/Day1 and Week 8</li> </ul> |
| Study Design | This is a Prospective, Vehicle Controlled, Double Blind, Multicenter, Randomized Phase II trial, comparing the effect of twice daily B244 application for 8 weeks vs. vehicle application on treatment of mild to moderate rosacea. |
| | <ul> <li>We will enroll approximately 130 subjects and complete 104 subjects.</li> <li>At Screening and Baseline: <ul> <li>All subjects must have diagnosis of mild to moderate Rosacea.</li> <li>Subjects must have IGA score of 2-3 and CEA score of 2-3 to qualify for the study.</li> </ul> </li> <li>After screening and recruitment, participants will be randomized to active or vehicle application for 8 weeks.</li> <li>Subjects will apply a total of 4 pumps of IP per application to the face twice-a-day</li> <li>Randomization will be 1:1 B244 to Vehicle.</li> <li>Subjects will be provided with cleanser and moisturizer to use for the duration of the study</li> <li>All B244 randomized subjects will be treated at the dose of 4x10° cells/ml via spray application</li> <li>Screening period will occur at Days -21 to -1</li> <li>Washout will occur after Screening visit (Days - 14 to -1)</li> <li>Randomization will occur during the baseline visit for the study Efficacy will be assessed using Investigator Global Assessment (IGA) score, Clinician's Erythema Assessment (CEA) score, Patient Self-Assessment (PSA) score and patient reported Skindex 16.</li> <li>Clinical assessments of response to treatment will be made at Week 1(Day 7), Week 4 (Day 28), and Week 8 (Day 56)</li> <li>At Baseline visit, subjects will receive a kit containing the drug product. Each bottle will be used for 2 weeks. At Week 4, subjects will return the used bottles from the kit and will be issued a new kit of drug product to be used from Week 4 through Week 8.</li> </ul> |

Subjects will stop applying investigational product at Week 8 and will return investigational product at that visit.





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN Version 2 Confidential 02-Apr-19 Subjects will come back for a 4-week posttreatment follow up visit at Week 12 (Day 84). Participant's safety will be monitored throughout the study. Safety will be assessed by monitoring reported adverse events, vital signs, clinical chemistry and hematology and overall tolerability of the investigational product. Subjects would be required to discontinue the investigational product under the following circumstances: o Development of an intercurrent illness that would jeopardize the safety, or significantly affect assessments of clinical status of a subject Either at the discretion of the Investigator or at the participant's request o Development of any investigational product-related SAE Suspected or laboratory-confirmed pregnancy Number of Approximately 130 subjects are planned to be enrolled, and assuming a **Subjects and Sites** 20% drop out rate, the planned overall sample size for this clinical trial is approximately 104 adult male and female subjects, 18 years of age and older with mild to moderate rosacea. Subjects will be randomized at a 1:1 ratio (B244: vehicle) at about 8 clinical research centers in the United States. INCLUSION CRITERIA **Eligibility Criteria** 8. Aale a n d female subjects A clinical diagnosis of mild to moderate facial rosacea. In good general health as determined by a thorough medical history, physical examination, clinical chemistry and hematology. A Clinician Erythema Assessment (CEA) score of 2-3 at Screening and at Baseline Visits (prior to the investigational product application). Mild to Moderate IGA score of 2-3 at Screening and at Baseline Visits (prior to the investigational product application). Willing to refrain from using any topical or systemic treatments for the treatment of rosacea, other than the investigational product. Females of childbearing potential with a negative urine pregnancy test (UPT) at Screening and Baseline/Day 1 (prior to the investigational product application).

Ability to comprehend and comply with study procedures. Agree to commit to participate in the current protocol.





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN Version 2

Provide written informed consent prior to any study procedure being performed.

#### **EXCLUSION CRITERIA**

Any subject who meet one or more of the following criteria are excluded from this study.

- Female subjects who are pregnant, lactating or who are trying to conceive will be excluded from participation in this study.
- Any uncontrolled chronic or serious disease or medical condition that would normally prevent participation in a clinical trial, or, in the judgment of the Investigator, would put the subject at undue risk, or might confound the study assessments (e.g., other dermatological diseases), or might interfere with the subject's participation in the study, (e.g., planned hospitalization during the study).
- Particular forms of rosacea (e.g., rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin, Ocular rosacea Phymatous rosacea, Steroid-induced rosacea, severe rosacea including pyoderma faciale) or other concomitant facial dermatoses that are similar to rosacea such as peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus, or actinic telangiectasia.
- Presence of three (3) or more facial inflammatory lesions of rosacea
- Any skin condition which in the investigator's opinion may interfere with the evaluation of rosacea.
- Severe papulopustular rosacea requiring systemic treatment.
- Participation at the time of eligibility assessment (Screening) in any other investigational drug or device study or may have participated within 30 days prior to Screening.
- Commencement of new hormonal therapy or dose change to hormonal therapy within 90 days prior to baseline. Dose and frequency of use of any hormonal therapy started more than 90 days prior to baseline must remain unchanged throughout the study. Hormonal therapies include, but are not limited to, oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (e.g. vaginal ring or transdermal hormone contraception).






- Presence of beard or excessive facial hair at Screening which would interfere with the study treatments or study assessments and refusal to remove for duration of study.
- Current treatment with monoamine oxidase (MAO) inhibitors, barbiturates, opiates, sedatives, systemic anesthetics, or alphaagonists.
- Carcinoid, Pheochromocytoma or other systemic causes of flushing.
- Known sensitivity to B244 or its components.
- Refusal to submit to blood and urine sampling for laboratory analysis.
- Treatment with the following:

**Prohibited Topical Treatments:** 

| Topical Treatment | Prohibited Time |
|------------------------------------------|-----------------|
| Topical Treatment | |
| | Frame prior to |
| A | Baseline |
| Astringents or abrasives | 2 days |
| RHOFADE™ (oxymetazoline HCl) Cream,1% | 1 week |
| Bleach baths | 1 week |
| Mirvaso (brimonidine) topical cream | 1 week |
| Vinegar | 1 week |
| Topical Prescription/OTC medications for | 1 week |
| treatment of acne | |
| Soolantra (Ivermectin 1%) topical cream | 1 week |
| Topical Antibiotic | 2 weeks |
| Use of over the counter antimicrobial | 2 weeks |
| Benzoyl Peroxide | 2 weeks |
| Immunomodulators | 4 weeks |
| Oracea (doxycycline) topical cream | 2 weeks |
| Corticosteroids | 4 weeks |
| Electrocoagulation, Dermabrasion; Facial | 4 weeks |
| peels | |
| Dermatologic/surgical procedure on the | 4 weeks |
| face | |
| Topical Prescription medications for the | 4 weeks |
| treatment of rosacea (e.g. azelaic acid, | |
| metronidazole, etc.) | |
| Laser, Phototherapy, Photodynamic | 4 weeks |
| Therapy or IPL (intense pulsed light) | |
| treatment | |
| treatment | |






|---|---|---|
| | Prescription or over the counter topical retinoid use on the face (e.g., tretinoin, tazarotene, adapalene) | 4 weeks |
| | Prohibited Systemic Treatments: | |
| | Topical Treatment | Prohibited Time Frame prior to Baseline |
| | Exposed to excessive ultraviolet (UV) radiation and/or subject was unwilling to refrain from excessive exposure to UV radiation during the course of the study. | 1 week |
| | Prescription anti inflammatory Prescription/OTC anti-inflammatory | 2 weeks 2 weeks |
| | medications (excludes low dose aspirin) Systemic Antibiotics | 4 weeks |
| | Prescription medications for the treatment of rosacea (e.g. doxycycline, tetracycline, macrolides) | 4 weeks |
| | Prescription medications for treatment of acne | 4 weeks |
| | Corticosteroids (oral or injectable) | 4 weeks |
| | Immunomodulators Oral retinoid use (e.g., isotretinoin), vitamin A supplements greater than 10,000 units/day | 12 weeks 6 months |
| Withdrawal and<br>Early<br>Discontinuation | A subject may voluntarily withdraw from the study at any time and for any reason without prejudice to his or her future medical care. The Investigator, Sponsor, or Medical Monitor may also withdraw a subject at any time if it is medically necessary or in the interest of subject's safety. If a subject discontinues prematurely, the Investigator will perform Early Termination (ET) visit, capturing the reason for discontinuation. Further details are provided in section 5.2 & 5.3 of the Protocol RB244-001 v4.0. | |
| Prohibited<br>Concomitant<br>Medication | Prohibited Therapies are those medicinal products and treatment methods that are not allowed during the study period and within the timeframes specified in the section 8.1 of the Protocol RB244-001 v 4.0. | |
| Study Drug | Study drug includes Test and Placebo drug procupility study drug as matching 30ml/bottle, lab Test Drug: B244, 30ml/bottle (AOBion | peled for a blinded study. |
| | Placebo: Vehicle, 30ml/bottle (AOBio | |






|---|---|
| Duration of Patient<br>Study Participation | Up to $84 \pm 2$ days |
| Study Endpoints | PRIMARY |
| | <ul> <li>The primary safety endpoint is to assess the safety and<br/>tolerability of B244 applied twice daily (BID) to the face for 8<br/>weeks in subjects with mild to moderate rosacea based on the<br/>number of AE &amp; SAE.</li> </ul> |
| | EXPLORATORY |
| | To assess the efficacy of B244 in subjects with mild to moderate rosacea. |
| | <ul> <li>Change of IGA score at Baseline to Week 1, Week 4, Week 8<br/>and Week 12</li> </ul> |
| | <ul> <li>Change of CEA score at Baseline to Week 1, Week 4, Week 8<br/>and Week 12.</li> </ul> |
| | <ul> <li>Change of PSA score at Baseline to Week 1, Week 4, Week 8 and Week 12.</li> <li>Change of Skindex 16 patient reported outcome from Baseline to Week 1, Week 4, Week 8 and Week 12</li> </ul> |
| | • IGA treatment success, defined as "clear" or "almost clear" with a 2-grade improvement in IGA score from baseline to the end of treatment. |
| | CEA treatment success, defined as "clear" or "almost clear" with a 2-grade improvement in CEA score from baseline to the end of treatment |
| Statistical Analysis | SAFETY ANALYSIS |
| | The reporting of safety data is descriptive (arithmetic mean, standard deviation (SD), coefficient of variation (CV), median, minimum, and maximum) will be calculated for quantitative safety data as well as for the difference from baseline, when appropriate. |
| | The analysis will include all subjects who receive at least one dose of investigational product. The variables for safety endpoints are AEs, Local Application Site Reactions, vital signs measurements, clinical chemistry and hematology. AEs will be summarized based on the frequency of AEs and their severity for all treated subjects. All AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA) and summarized by treatment group. Data will be summarized using preferred term and primary system organ class, including verbatim term, dose level, severity, and relationship to treatment, will be provided. |






Concomitant medications will be listed by treatment and coded using the most recent version of the World Health Organization (WHO) Drug Dictionary (DD).

#### **EFFICACY ANALYSIS**

The Evaluable Period for the outcome variables will be weeks 1, 4, 8 and 12. The superiority of the drug over the vehicle will be tested at week 8 based on the probability of improvement from baseline with a continuity-corrected Z-tests comparing the change from baseline of treatments vs Placebo. For all other evaluable periods, descriptive statistics for the change from baseline will be shown.

The change from baseline score of Skindex-16 will be compared among treatments at Week 12 using an ANOVA.






#### STATISTICAL ANALYSIS PLAN

Version 2 02-Apr-19

### **Table of Contents**

## Contents

| S | TATIS: | ΓΙCAL ANALYSIS PLAN REVIEW AND APPROVAL | 2 |
|---|---|---|---|
| ΡI | котос | OL SYNOPSIS | 3 |
| 1 | LIST | OF ABBREVIATION | 14 |
| 2 | INT | RODUCTION | 16 |
| | 2.1 | Study Overview | 16 |
| | 2.2 | Study Flowchart | 18 |
| | 2.3 | Schedule of Activities | 19 |
| 3 | STU | DY OBJECTIVE AND ENDPOINTS | 21 |
| | 3.1 | Study Objectives | 21 |
| | 3.1. | 1 Primary Objective | 21 |
| | 3.1. | 2 Exploratory Objectives | 21 |
| | 3.2 | Study Endpoints | 21 |
| | 3.2. | Safety & Tolerability (Primary) | 21 |
| | 3.2. | 2 Efficacy (Exploratory) | 21 |
| 4 | STU | DY DESIGN | 22 |
| | 4.1 | Summary of Study Design | 22 |
| | 4.2 | Definition of Study Drugs | 22 |
| | 4.3 | Sample Size Considerations | 23 |
| | 4.4 | Study Withdrawal | 23 |
| | 4.5 | Early Discontinuation | 24 |
| 5 | PLA | NNED ANALYSIS | 24 |
| | 5.1 | Final Analysis | 24 |
| 6 | GEN | IERAL CONSIDERATION FOR DATA ANALYSIS AND HANDLING | 24 |
| | 6.1 | General Summary Table and Individual Subject Data Listing | 24 |
| | 6.2 | General Summary Table and Individual Subject Data Listing Considerations | 25 |
| | 6.3 | Data Management | 26 |
| | 6.4 | Data Presentation Conventions | 26 |
| | 6.5 | Analysis Populations | 27 |
| | 6.5. | 1 Screen Failures | 27 |





| Protocol: RE Confidential | | Version 2<br>02-Apr-19 |
|---|---|---|
| 6.5.2 | Safety Population | |
| 6.5.3 | mITT Population | 27 |
| 6.5.4 | Per-Protocol (PP) Population | 27 |
| 6.6 Ba | seline Definition | 28 |
| 6.7 De | rived and Transformed Data | 28 |
| 6.7.1 | Baseline Age | 28 |
| 6.7.2 | Study Day | 28 |
| 6.7.3 | Multiple Assessments | 28 |
| 6.7.4 | Handling of Missing Data & Sensitivity Analysis | 28 |
| 6.7.5 | Missing Start and Stop Dates for Prior and Concomitant Medication | 29 |
| 6.7.6 | Safety Parameters | 29 |
| 6.7.7 | Missing Start and Stop Dates for Adverse Events | 29 |
| 7 DATA A | NALYSES | 31 |
| 7.1 Su | bjects Disposition | 31 |
| 7.2 Pr | otocol Deviations | 31 |
| 7.3 De | mographic and Baseline Characteristics | 32 |
| 7.4 Stu | udy Drug Exposure | 32 |
| 7.5 M | edical History | 32 |
| 7.6 Co | ncomitant Medication | 33 |
| 7.7 Vit | al Signs and Physical Examination | 33 |
| 7.8 La | boratory Data | 33 |
| 7.9 Vis | sit Windows | 33 |
| 8 STATIST | TICAL ANALYSES | 33 |
| 8.1 Sa | mple Size Determination | 33 |
| 8.2 Sa | fety Analysis | 34 |
| 8.2.1 | Primary Safety Endpoint | 34 |
| 8.3 Eff | icacy Analysis | 34 |
| 8.4 Se | nsitivity Analysis | 35 |
| 9 REFERE | NCES | 36 |
| 10 APPE | NDIX | 37 |
| 10.1 AP | PENDIX A: Tables | 37 |
| 10.1.1 | General | 37 |





| Protocol: RB2<br>Confidential | 244-001 | STATISTICAL ANALYSIS PLAN | Version 2<br>02-Apr-19 |
|---|---|---|---|
| 10.1.2 | Efficacy | | 49 |
| 10.1.3 | Safety | | 53 |
| 10.2 APP | ENDIX B: Listings | | 57 |
| 10 3 ΔΡΡ | FNDIX C. Figures | | 5.2 |






### 1 LIST OF ABBREVIATION

| Abbreviation | Full Form |
|--------------|------------------------------------------------|
| AE | Adverse Event |
| AOB | Ammonia-Oxidizing Bacteria |
| BID | Bis in Die (twice a day) |
| BP | Blood Pressure |
| CEA | Clinician Erythema Assessment |
| CRA | Clinical Research Associate |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CTMF | Clinical Trial Master File |
| CTP | Clinical Trial Protocol |
| eCRF | Electronic Case Report Form |
| EOS | End of Study |
| ET | Early Termination |
| ETR | Erythematotelangiectatic rosacea |
| GCP | Good Clinical Practice |
| IB | Investigator's Brochure |
| ICH | International Conference On Harmonization |
| IEC | Independent Ethics Committee |
| IGA | Investigator Global Assessment |
| IGE | Investigator's Global Evaluation |
| IP | Investigational Product |
| IPL | Intense Pulsed Light |
| IRB | Institutional Review Board |
| ISF | Investigator Site File |
| IUD | Intrauterine Device |
| IUS | Intrauterine system |
| IWRS | Interactive Web Response System |
| LOCF | Last Observation Carried Forward |
| mITT | Modified Intent-To-Treat |
| NSAID | Nonsteroidal Anti-inflammatory Drug |
| OTC | Over the Counter |
| PP | Per-Protocol |
| PRN | Pro Re Nada (as needed) |
| PRN | Pro Re Nada (as needed) |
| PSA | Patient Self-Assessment |
| RR | Relative Risk |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SI | Simple Imputation |
| SOP | Standard Operating Procedures |
| SUSAR | Suspected Unexpected Serious Adverse Reactions |
| TEAE | Treatment Emergent Adverse Event |




Protocol: RB244-001 STATISTICAL ANALYSIS PLAN Version 2 Confidential 02-Apr-19

Upper Limit of Normal Range Urine Pregnancy Test Ultraviolet ULN

UPT

UV

White Blood Cell Count WBC





### 2 INTRODUCTION

This document describes the statistical methods and data presentations to be used in the summary and analysis of data from Protocol RB244-001. Background information is provided for the overall study design and objectives. The reader is referred to the study protocol and electronic case report forms (eCRFs) for details of study conduct and data collection.

# 2.1 Study Overview

The proposed study is aimed to evaluate the safety and efficacy of B244 topical spray. A Vehicle-Controlled, Double-Blind, Multicenter, Randomized Study Design has been Selected to Evaluate the Safety and Efficacy of the B244 Investigational product in the Treatment of Mild-to-Moderate Rosacea.

There is no cure for rosacea and treatment is aimed at alleviating the symptoms. Topical or oral medications are generally prescribed for mild to moderate papulopustular rosacea. These topical medications include: metronidazole, azelaic acid, sodium sulfacetamide and sulfur, erythromycin, and tretinoin8. Currently these approved topical medications may cause local irritation to the skin. The oral medications prescribed for severe disease include tetracycline, doxycycline, minocycline, erythromycin and metronidazole. The systemic therapies may result in systemic adverse events such as gastrointestinal upset and photosensitivity.

It is believed, that topical application of Ammonia-Oxidizing Bacteria (AOB) will reduce survival of pathogenic bacteria present on the skin and thus improve rosacea symptoms in those affected by it. B244 is being developed as a 'live topical' to provide a natural source of AOB and NO/NO2 to the human skin.

This is a Prospective, Vehicle Controlled, Double Blind, Multicenter, Randomized Phase II trial, Comparing the effect of twice daily B244 application for 8 weeks vs. vehicle application on treatment of mild to moderate rosacea. At Screening and Baseline all subjects must have clinical diagnosis of mild to moderate rosacea and subjects must have IGA score of 2-3 and CEA score of 2-3 to qualify for the study.

After screening and recruitment, participants will be randomized to active or vehicle application for 8 weeks. Subjects will apply a total of 4 pumps of IP per application to the face twice-a-day. Subjects will be provided with cleanser and moisturizer to use for the duration of the study. All B244 randomized subjects will be treated at the dose of  $4 \times 10^9$  cells/ml via spray application.

Efficacy will be assessed using Investigator Global Assessment (IGA) score, Clinician's Erythema Assessment (CEA) score, Patient Self-Assessment (PSA) score and patient reported Skindex 16. Participant's safety will be monitored throughout the study. Safety







will be assessed by monitoring reported adverse events, vital signs, clinical chemistry and hematology and overall tolerability of the investigational product.

Approximately 130 subjects are planned to be enrolled, and assuming a 20% drop out rate, the planned overall sample size for this clinical trial is approximately 104 adult male and female subjects, 18 years of age and older with mild to moderate rosacea. Subjects will be randomized at a 1:1 ratio (B244: Vehicle) at about 8 clinical research centers in the United States.

The entire study will consist of a total of 6 visits:

- Visit 1(Day -21 to -1): Screening will occur at Days -21 to -1, followed by Washout (Days -14 to -1).
- Visit 2(Baseline/ Day 1): Randomization will occur during the baseline visit for the study (Day 1).
- Visit 3 5(Day 7 ± 2 [Week 1], Day 28 ± 2 [Week 4], Day 56 ± 2 [Week 8]): Clinical assessments of response to treatment will be made at Week 1(Day 7), Week 4 (Day 28), and Week 8 (Day 56).
- Visit  $6(\text{Day }84 \pm 2)$ : Subjects will come back for a 4-week post-treatment follow up visit at Week 12 (Day 84).





STATISTICAL ANALYSIS PLAN Protocol: RB244-001


#### 2.2 **Study Flowchart**

Figure 1. Study Flowchart

### STUDY SCHEMA









# 2.3 Schedule of Activities

Table 1: Schedule of Study Activities

| Visit Name | Screening | Baseline/<br>DAY 1 | Week<br>1 | Week 4 | Week 8 | Week 12/<br>End of<br>Study Visit | Early<br>Termination<br>Visit |
|---|---|---|---|---|---|---|---|
| Visit number | Visit 1 | Visit 2 | Visit<br>3 | Visit 4 | Visit 5 | Visit 6 | |
| Visit window in days | -21 to -1 | 1 | 7+/-2 | 28 +/- 2 | 56 +/- 2 | 84 +/- 2 | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | X | | | | | |
| Demographics | X | | | | | | |
| Medical History | X | X | | | | | |
| Concomitant Medications | X | X | X | X | X | X | X |
| Physical Exam | X | X | | | | X | X |
| BP & Pulse <sup>2</sup> | X | X | X | X | X | X | X |
| Urine pregnancy test for WOCBP <sup>1</sup> | X | X | X | X | X | X | X |
| Clinical chemistry and hematology and urinalysis <sup>3</sup> | X | X | | X | X | | X |
| Biomarkers <sup>4</sup> | | X | | | X | | X |
| CEA | X | X | X | X | X | X | X |
| IGA | X | X | X | X | X | X | X |
| Skindex 16 | X | X | X | X | X | X | X |
| PSA score | X | X | X | X | X | X | X |
| Telangiectasia Evaluation | | X | | | X | | X |
| Fitzpatrick skin type | X | | | | | | |
| IWRS | | X | | X | | | |
| Dispense Investigational product to Subject 5/6 | | X | | X | | | |
| Collect Investigational product from Subject <sup>5</sup> | | | | X | X | | X |





#### 1. DD244 001 CTATICTICAL ANIALYCIC DLAN


| Visit Name | Screening | Baseline/<br>DAY 1 | Week<br>1 | Week 4 | Week 8 | Week 12/<br>End of<br>Study Visit | Early<br>Termination<br>Visit |
|---|---|---|---|---|---|---|---|
| Visit number | Visit 1 | Visit 2 | Visit<br>3 | Visit 4 | Visit 5 | Visit 6 | |
| Visit window in days | -21 to -1 | 1 | 7+/-2 | 28 +/- 2 | 56 +/- 2 | 84 +/- 2 | |
| Investigational product<br>Compliance <sup>5</sup> | | X | | X | X | | X |
| Study Cleanser and moisturizer dispensation <sup>9</sup> | | X | | X | | | |
| Study Cleanser and moisturizer collection | | | | | X | | X |
| Study Diary <sup>8</sup> | | X | X | X | X | | X |
| Study Counseling <sup>7</sup> | | X | X | X | X | | |
| AE Collection and<br>Assessment | X | X | X | X | X | X | X |

- 1. Urine pregnancy test for WOCBP will be done at every visit.
- 2. Blood pressure readings will be obtained at every visit. Subject should be allowed to rest for more than 5 minutes sitting, then BP measurements and pulse (x3) will be performed, using the non-dominant arm with a calibrated electronic sphygmomanometer. The average of the second and third readings will be documented.
- 3. Subjects should fast for at least 8 hours before the test. Laboratory work includes: hematology and Lipid Panel, Albumin, Alkaline Phos, ALT, AST, Total Bilirubin, BUN, BUN: Creatinine ratio, Calcium, Chloride, Creatinine, eGFR, Glucose, Potassium, Sodium, Uric Acid, and urinalysis. HIV Ab, HCV Ab, HBsAg. will only be done at screening.
- 4. Subjects should fast for at least 8 hours before the test.
- 5. Weight of the investigational product kit will be obtained at the Baseline visit. Study staff will be asked to weigh all dispensed bottles without the carton box PRE- FIRST DOSE. Weight will be recorded in grams.
- 6. Subjects will be asked to bring all dispensed bottles back for the Week 4 and Week 8 visits. Upon return for the study visit, all bottles will be weighed again without the carton box. Subjects will be asked to apply the investigational product twice daily. First investigational product application will happen at the site under medical supervision.
- 7. Subjects will be counseled on the use of study medication and answer any questions subject may have.
- 8. Subjects will be asked to fill out study diary for the duration of the study.
- 9. Cleanser and moisturizer will be dispensed at the Baseline visit. Subjects will be asked to refrain, if possible, from using any other cleanser and/or moisturizer on their face and apply the provided product while they are participating in the trial. Any leftover moisturizer /cleanser will be collected at Week 8 visit, at which point subjects will be asked to go back to their regular routine.





### 3 STUDY OBJECTIVE AND ENDPOINTS

### 3.1 Study Objectives

### 3.1.1 Primary Objective

To assess the safety and tolerability of B244 applied twice daily (BID) to the face for 8 weeks in subjects with mild to moderate rosacea.

### 3.1.2 Exploratory Objectives

To assess the efficacy of B244 in subjects with mild to moderate rosacea.

- o Proportion of subjects with IGA improvement at Week 8 relative to baseline.
- o Proportion of subjects with CEA improvement at Week 8 relative to baseline.
- o Change in IGA score from Baseline to Week 8.
- o Change in CEA score from Baseline to Week 8.
- o Proportion of Subjects with improvement in IGA or CEA at Week 1, Week 4, and Week 12.
- Change in Skindex 16 patient reported outcome from Baseline to Week 1, Week 4, Week 8, and Week 12.
- o Proportion of subjects with change in PSA at Week 1, Week 4, Week 8 and Week 12 from Baseline.
- Evaluation of Telangiectasia Score at Baseline/Day 1 and Week 8

# 3.2 Study Endpoints

### 3.2.1 Safety & Tolerability (Primary)

Safety and tolerability endpoints will consist of all adverse events reported during the study duration.

### 3.2.2 Efficacy (Exploratory)

- o Change of IGA score at Baseline to Week 1, Week 4, Week 8 and Week 12.
- o Change of CEA score at Baseline to Week 1, Week 4, Week 8 and Week 12.
- o Change of PSA score at Baseline to Week 1, Week 4, Week 8 and Week 12.
- Change of Skindex 16 patient reported outcome from Baseline to Week 1, Week 4, Week 8 and Week 12.
- o IGA treatment success, defined as "clear" or "almost clear" with a 2-grade improvement in IGA score from baseline to the end of treatment.
- o CEA treatment success, defined as "clear" or "almost clear" with a 2-grade improvement in CEA score from baseline to the end of treatment.





### 4 STUDY DESIGN

### 4.1 Summary of Study Design

This is a Prospective, Vehicle Controlled, Double Blind, Multicenter, Randomized Phase II trial, Comparing the effect of twice daily B244 application for 8 weeks vs. vehicle application on treatment of mild to moderate rosacea. We will enroll approximately 130 subjects and complete 104 subjects.

At Screening and Baseline, all subjects must have clinical diagnosis of mild to moderate rosacea and must have IGA score of 2-3 and CEA score of 2-3 to qualify for the study. After screening and recruitment, participants will be randomized to active or vehicle application for 8 weeks. Subjects will apply a total of 4 pumps of IP per application to the face twice-a-day. Randomization will be 1:1 B244 to Vehicle. Subjects will be provided with cleanser and moisturizer to use for the duration of the study. All B244 randomized subjects will be treated at the dose of  $4x10^9$  cells/ml via spray application. Screening will occur at Days -21 to -1. Washout will occur after Screening visit (Days -14 to -1) and randomization will occur during the baseline visit for the study (Day 1).

Efficacy will be assessed using Investigator Global Assessment (IGA) score, Clinician's Erythema Assessment (CEA) score, Patient Self-Assessment (PSA) score and patient reported Skindex 16. Clinical assessments of response to treatment will be made at Week 1(Day 7), Week 4 (Day 28), and Week 8 (Day 56). At Baseline visit, subjects will receive a kit containing the drug product. Each bottle will be used for 2 weeks. At Week 4, subjects will return the used bottles from the kit and will be issued a new kit of drug product to be used from Week 4 through Week 8. Subjects will stop applying investigational product at Week 8 and will return investigational product at that visit. Subjects will come back for a 4-week post-treatment follow up visit at Week 12 (Day 84). Participant's safety will be monitored throughout the study. Safety will be assessed by monitoring reported adverse events, vital signs, clinical chemistry and hematology and overall tolerability of the investigational product.

Subjects would be required to discontinue the investigational product under the following circumstances:

- Development of an intercurrent illness that would jeopardize the safety, or significantly affect assessments of clinical status of a subject
- Either at the discretion of the Investigator or at the participant's request
- Development of any investigational product-related SAE
- Suspected or laboratory-confirmed pregnancy

### 4.2 Definition of Study Drugs

Study drug includes Test and Placebo drug products. The Sponsor will supply study drug as matching 30ml/bottle, labeled for a blinded study.






Test Drug: B244, 30ml/bottle (AOBiome, LLC)
Placebo: Vehicle, 30ml/bottle (AOBiome, LLC)

### 4.3 Sample Size Considerations

Approximately 130 subjects are planned to be enrolled, and assuming a 20% drop out rate, the planned overall sample size for this clinical trial is approximately 104 adult male and female subjects, 18 years of age and older with mild to moderate rosacea. Subjects will be randomized at a 1:1 ratio (B244: Vehicle) at about 9 clinical research centers in the United States.

# 4.4 Study Withdrawal

A subject may voluntarily withdraw from the study at any time and for any reason without prejudice to his or her future medical care. The Investigator, Sponsor, or Medical Monitor may also withdraw a subject at any time if it is medically necessary or in the interest of subject's safety. Additional reasons for premature discontinuation of investigational product may include adverse events and major non-compliance with study procedures, as described below. The withdrawal of a subject from investigational product by the Investigator will be discussed with the Medical Monitor before the subject stops investigational product, whenever possible.

A subject will be discontinued from this study if any of the following criteria are met:

- Withdrawal of consent by the subject is received.
- In the opinion of the Investigator, Medical Monitor or Sponsor, it is not in the subject's best interests to continue in the study.
- Significant non-compliance with study procedures that would interfere with the study results or increase the subject's risks in the study, as determined by the Investigator.
- Development of an intercurrent illness that would jeopardize the safety, or significantly affect assessments of clinical status of a subject.
- Development of any investigational product-related SAE.
- Suspected or laboratory-confirmed pregnancy.

Subjects who discontinued early from the study due to lack of treatment effect after completing at least four weeks of treatment (Day 28) will be included in the mITT and PP population as treatment failures and the change in IGA and CEA from the baseline visit to the last completed visit prior to discontinuation due to lack of efficacy will be carried forward in the primary endpoint analysis. Subjects discontinued early for other reasons will be excluded from the PP population.





### 4.5 Early Discontinuation

CLINICAL RESEARCH OPTIMIZED™

If a subject discontinues prematurely, the Investigator will perform Early Termination (ET) visit, capturing the reason for discontinuation.

If a subject does not return for a scheduled visit, every effort will be made to contact the subject and document the End of Study visit assessments. The Investigator must document the primary reason for discontinuation of a study subject in the source document and on the appropriate electronic case report form (eCRF).

### 5 PLANNED ANALYSIS

### 5.1 Final Analysis

Final analysis is planned for the study after the database lock. The final analysis will follow instructions presented in this SAP.

# 6 GENERAL CONSIDERATION FOR DATA ANALYSIS AND HANDLING

### 6.1 General Summary Table and Individual Subject Data Listing

Summary tables and listings (e.g., post text tables and individual subject data listings are prepared according to ICH Guideline E3) include a "footer" providing explanatory notes that indicate as a minimum:

- SAS program name.
- Programmer.
- Date of data extraction.
- Date of output generation.

Post text tables also include reference(s) to the subject data listing(s) that supports the summary data. The data extraction date links the output to the archived database that is locked to ensure the replication of the results.

Post text tables will be organized with respect to treatment group and a column will be included to summarize all treated subjects. The order of drug presentation will be investigational drug first followed by the vehicle control. A total column will appear as the last column. The summary tables clearly indicate the number of subjects to which the data apply and unknown or not performed are distinguished from missing data.

Summary tables for medications and medical conditions are coded according the WHO Drug Dictionary. Adverse event preferred terms and body/organ systems are coded using





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN


the MedDRA dictionary. The MedDRA dictionary can be used, as well, in the coding of signs and symptoms, medical history, physical examination abnormalities, and clinical diagnoses.

Supportive individual subject data listings, as a minimum, are sorted and presented by treatment group and subject id. Listings also include visit number, visit date, and days relative to the initiation of double-blind treatment.

#### 6.2 General Summary Table and Individual Subject Data Listing **Considerations**

The default convention is to number tables and listings using a decimal system to reflect main levels of unique tables and listings and sub-levels of replicate tables and listings with two digits per level (e.g., Table XX.YY.ZZ. ...).

- The first level number should be consistent with the corresponding CSR appendix in which the tables or listings will appear. For example, the post text tables usually occupy Appendix 14 and the individual subject data listings are put in Appendix 16. All post text tables should have a main number level 14 and listings 16. The subject accounting and disposition table is usually first in the first section of the report and should be numbered Table 14.1. The supportive subject data listing would be Listing 16.1. A subset by sex 2. Subject accounting and final disposition should appear as the second level number (Table 14.1 series). Baseline and demographic profile occupy the next sub-level (Table 14.2 series). Efficacy should come next (Table 14.3 series) followed by safety Table 14.4 series). Reasons for subjects' being excluded from efficacy and protocol violation summary tables should appear as the last level (Table 14.5 series). Similar conventions should be applied to the subject data listings.
- The title should be complete, accurate, and concise. The last line of the title should provide the analysis group being summarized (e.g., Intent-to-Treat Subjects or Per-Protocol Efficacy Subjects). If possible, the units of measurement for data contained in the table can appear in parentheses to conserve space in the body of the table. For example, the summary of vital signs title could read "Summary of Sitting and Standing Blood Pressure (mmHg) and Heart Rate (bpm)." Whether in the title or body of a table or listing, units must always be specified for all appropriate data.
- If possible, variables being summarized, and statistics reported should appear in the left most column of a table. The next columns for treatment groups should report the data from left to right for the investigational drug, placebo, comparative agents, and (optional) all treated subjects, respectively.

In general, the listings should be sorted and presented by treatment assignment, investigational site, and subject number. Treatment assignment and site can appear in the banner of the listing. From left to right, the subject number, visit number, visit date, and relative day should appear.





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN


All tables and listings must have explanatory notes that give, as a minimum, data extraction date, output generation date, complete program name and path where it is stored, as appropriate. The definition of all derived variables and decodes for coded data must appear in the notes. Due to space limitations, tables and listings may require a page of notes as a one-time preface to the output.

#### 6.3 **Data Management**

Biorasi will create SDTM data sets and ADaM analysis data sets using (SAS®) software. Data analyses and summary tables are generated using SAS version 9.4 or above

#### 6.4 **Data Presentation Conventions**

Continuous variables (e.g. age) are summarized using descriptive statistics (the number of subjects with available data, the mean, standard deviation (SD), median, minimum and maximum). Categorical variables (e.g. race) are summarized using counts and percentages. Percentages are calculated using the total subjects per treatment group.

The following conventions are applied to all data presentations and summaries:

- For continuous variables, all mean and median values are formatted to one more decimal place than the measured value. Standard deviation values are formatted to two more decimal places than the measured value. Minimum and maximum values are presented with the same number of decimal places as the measured value.
- For categorical variables, the number and percentage of responses are presented in the form XX (XX.X %) where the percentage is in the parentheses.
- Date variables are formatted as DDMMMYYYY for presentation. Time is formatted in military time as HH:MM for presentation.
- Wherever possible, data will be decimal aligned.
- P-values, if applicable, will be presented to 4 decimal places. If the p-value is less than 0.0001 then it will be presented as < 0.0001.

Unless otherwise stated, any statistical tests performed will use 2-sided tests at the 5% significance level.

The table and listing shells and table of contents as part of this SAP provide the expected layout and titles of the tables, listings and figures. Any changes to format, layout, titles, numbering, or any other minor deviation will not necessitate a revision to the SAP nor will it be considered a deviation from planned analyses. Only true differences in the analysis methods or data handling will necessitate such documentation. The appropriate listings supporting the tables will be included and are not specified in the individual sections throughout the document.





### 6.5 Analysis Populations

### 6.5.1 Screen Failures

Investigators must account for all subjects who sign informed consent and will maintain an Enrollment Log capturing subjects screened and indicating who was enrolled or excluded and the reason why. If the subject is found not to be eligible prior to enrollment, the reason(s) for ineligibility must be documented by the Investigator.

These subjects will neither contribute to data presentations nor be included in formal statistical analyses. The number of screen failures will be included in the data disposition table. Subject Numbers assigned to subjects who fail Screening will not be re-used.

### **6.5.2 Safety Population**

The safety population includes all randomized subjects who received investigational product.

### 6.5.3 mITT Population

A modified intent-to-treat population includes all subjects who are randomized, applied at least one dose of assigned product, and returned for at least one post-baseline evaluation visit.

### 6.5.4 Per-Protocol (PP) Population

The PP population includes all randomized subjects who met all inclusion/exclusion criteria, were compliant with the assigned study treatment, returned to the study site for the primary endpoint visit within the specified window ( $\pm 2$  days) OR discontinued from the study as a treatment failure, and did not have any major protocol violations.

Subjects who administered at least 50 % of IP, have at least one baseline and post baseline in clinic visit and did not have any major protocol violations.

Subjects who discontinued early from the study due to lack of treatment effect after completing at least eight weeks of treatment should be included in the mITT and PP population as treatment failures and the change in IGA and CEA from the baseline visit to the last completed visit prior to discontinuation due to lack of efficacy should be carried forward in the primary endpoint analysis. Subjects discontinued early for other reasons should be excluded from the PP population but included in the mITT population.

The results in the mITT population will be considered definitive for superiority of each active treatment to vehicle with those in the PP population considered supportive. Safety analyses will be performed using the Safety population.






### **6.6** Baseline Definition

The Baseline visit (Day 0) will take place once the results of Screening assessments are obtained, suggesting that the subject is eligible for entering the study. During this visit, those subjects who qualify for entering the study will be randomized to one of the study arms in a ratio of 1:1.

### 6.7 Derived and Transformed Data

### 6.7.1 Baseline Age

Subject's age in years will be calculated based on the date of the Baseline Visit date using the following formula:

Age (years) = FLOOR ((INTCK ('month', Date of Birth, Date of Baseline Visit) - (DAY(Date of Baseline Visit) < MIN(DAY(Date of Birth), DAY (INTNX ('month', Date of Baseline Visit, 1) - 1)) / 12); where:

- o FLOOR () is a SAS function that returns the largest integer that is less than or equal to the argument.
- o INTCK () is a SAS function that returns the number of interval boundaries of a given kind that lie between two dates, times, or datetime values.
- o DAY () is a SAS function that returns the day of the month from a SAS date value.
- o INTNX () is a SAS function that increments a date, time, or datetime value by a given time interval, and returns a date, time, or datetime value.

### 6.7.2 Study Day

Day 1 is defined as the day after the baseline when the subject will receive the first dose.

- For a visit date on or after the date of the first dose:
   Study Day = (date of interest date of first dose) + 1
- For a visit date before the date of the first dose:
   Study Day = (date of interest date of first dose)

### **6.7.3** Multiple Assessments

No multiple assessment for same visit are scheduled.

### 6.7.4 Handling of Missing Data & Sensitivity Analysis

For the primary and secondary analysis no missing values will be imputed. A sensitivity analysis will be performed by Multiple Imputation Regression Analysis using the following factors: treatment, age, gender, race, baseline IGA, baseline CEA, baseline PSA, smokers/non-smokers and the results of the same variable from previous visits.





STATISTICAL ANALYSIS PLAN

Protocol: RB244-001 Version 2 Confidential 02-Apr-19

### 6.7.5 Missing Start and Stop Dates for Prior and Concomitant Medication

#### Start date:

- o If start date is completely missing, start date will not be imputed.
- o If (year is present, and month and day are missing) or (year and day are present, and month is missing), set month and day to January 1.
- o If year and month are present and day is missing, set day to the 1st day of month

### Stop date:

- o If end date is completely missing, end date will not be imputed.
- o If (year is present, and month and day are missing) or (year and day are present, and month is missing), set month and day to December 31st.
- o If year and month are present and day is missing, set day to the last day of month.

### **6.7.6 Safety Parameters**

Safety and tolerability endpoints will consist of all adverse events (AEs) reported during the study duration from the date of randomization through Week 12 (End of Study Visit).

Specific AEs are defined below.

Treatment-Emergent Adverse Events (TEAE): Any AE with onset after the first dose of study medication through 56 days after the last dose of study medication.

Serious Adverse Event (SAE): An AE occurring at any dose that results in any of the following outcomes: death, a life-threatening AE, in-patient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect.

Associated with Use of the Study Drug: There is a reasonable possibility that the experience may have been caused by the study drug. If the Investigator does not know whether or not study drug caused the event, then the event will be handled as "related to study drug" for reporting purposes. The determination of whether an AE is related to study drug is as follows:

- Related: The AE has a missing, unknown, possible, probable or definite relationship to the study medication.
- Not related: The AE is unlikely or definitely unrelated to the study drug.

### 6.7.7 Missing Start and Stop Dates for Adverse Events

#### Start date:

o If start date is completely missing, start date is set to date of first dose.





#### STATISTICAL ANALYSIS PLAN

Protocol: RB244-001 Version 2 Confidential 02-Apr-19

> If (year is present, and month and day are missing) or (year and day are present, and month is missing):

> > If year = year of first dose, then set month and day to month and day of first dose.

If year < year of first dose, then set month and day to December 31st.

If year > year of first dose, then set month and day to January 1st.

If month and year are present and day is missing:

If vear = vear of first dose and

- If month = month of first dose, then set day to day of first dose
- If month < month of first dose, then set day to last day of month.
- If month > month of first dose, then set day to 1st day of month.

If year < year of first dose, then set day to last day of month.

If year > year of first dose, then set day to 1st day of month.

### Stop date:

If the outcome of the AE was ongoing or unknown, then the rules outlined below will not be applied.

- o If stop date is completely missing, stop date is set to date of study discontinuation.
- o If (year is present, and month and day are missing) or (year and day are present, and month is missing):

If year = year of study discontinuation, then set month and day to month and day of study discontinuation.

If year < year of study discontinuation, then set month and day to December 31st.

If year > year of study discontinuation, then set month and day to December 31st.

If month and year are present and day is missing:

If year = year of study discontinuation and

- If month = month of study discontinuation, then set day to day of study discontinuation date.
- If month < month of study discontinuation, then set day to last day of month.
- If month > month of study discontinuation, then set day to last day of month.

If year < year of study discontinuation, then set day to last day of month. If year > year of study discontinuation, then set day to last day of month.





# 7 DATA ANALYSES

The data analysis will be conducted on all participant data when the trial ends. Subjects will be pooled across all sites. Data will be presented by treatment group and overall. Categorical variables will be summarized by frequency distributions (number and percentages of subjects) and continuous variables will be summarized by descriptive statistics (mean, standard deviation, etc.).

Adverse events will be summarized by treatment group using the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment-emergent AEs (TEAEs), treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, discontinuations due to AEs, and AEs Grade 3 severity. By-subject listings will be provided for any deaths, SAEs, and AEs leading to discontinuation.

Descriptive statistics for each treatment group will be provided for clinical laboratory values (e.g., hematology, serum chemistry, and urinalysis) and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation. Abnormal clinical laboratory values will be listed.

All data will be provided in by-subject listings.

### 7.1 Subjects Disposition

The subject disposition summary will include the number screened, the number of screen failures, the number enrolled, the number in each patient population for analysis, the number who completed the study, the number who discontinued the study and reason for discontinuation from the study. Disposition data will be summarized by treatment and overall.

A by-subject data listing of study completion information including the reason for study discontinuation will be presented. A by-subject listing of inclusion/exclusion criteria not met will also be presented.

### 7.2 Protocol Deviations

A summary of all protocol deviations on ITT population by type will be generated. Protocol deviation data will be summarized by treatment and overall. A by-subject data listing of protocol deviations will also be presented.

All protocol deviations will be presented in a data listing.






### 7.3 Demographic and Baseline Characteristics

Demographic and baseline characteristic data summarization will be performed to descriptively assess the comparability of treatment groups. Data to be tabulated will include age, race, ethnicity, height, weight, and BMI, as well as baseline characteristics related to medical history, including hypertension, diabetes, smoking history.

### 7.4 Study Drug Exposure

At Baseline visit, Subjects will receive a kit containing (2) two 30 ml white bottles. Each bottle will be used for 2 weeks. At Week 4, subjects will return the used bottles from the kit and will be issued a new kit of two 30mL white bottles to be used from Week 4 through Week 8.

The cumulative amount of study drug exposure will be estimated by calculating the difference between the weight of the 2 bottles of drug at the time the drug was dispensed at Baseline/Week 4 and the weight of the 2 bottles at Week 4/Week 8. Differences will be summed together.

The amount of product used per day will be estimated by dividing the change by the number of days the subject was on treatment. These weights will be compared to the weight of the product that would be used if the subject was compliant with the protocol. Percent compliance will be calculated as follows:



The number of days the subject administered study drug, the amount of product used, and the percent compliance will be summarized by treatment group and presented in a by-subject data listing. The subject listing will also include by-visit IP weights. Percent compliance will be calculated only for subjects who returned the study drug at the end of the treatment. In the listing, subjects who withdrew from the study early will be flagged.

### 7.5 Medical History

A by subject data listing of medical history will be presented. Medical history will be coded using MedDRA v20.0, and the number and percentage of patients experiencing at least 1 such diagnosis by MedDRA System Organ Class (SOC) and preferred term (PT) will be reported.






### 7.6 Concomitant Medication

Concomitant medications will be coded using the World Health Organization (WHO) dictionary. Results will be tabulated by anatomic therapeutic class (ATC) and preferred term.

This data will be summarized by treatment group. Previous and concomitant medications will be presented in a data listing.

### 7.7 Vital Signs and Physical Examination

Vital sign measurements will be presented for each subject in a data listing. Systolic blood pressure, diastolic blood pressure, heart rate, and weight will be summarized as actual value and change from baseline by visit.

All physical examination findings will be presented in a data listing.

### 7.8 Laboratory Data

Clinical laboratory values will be expressed in SI units reported by the central laboratory.

The actual value and change from screening will be summarized for each clinical chemistry, hematology, lipid panel, HbA1C and urinalysis parameters and by each visit. In the event of repeat values, the last non-missing value per visit will be used.

Sample for Serology was collected only at Baseline. Hence Serology data will be only provided in a listing.

All laboratory data will be also provided in data listings. Values outside of the lab parameter's normal range will be flagged as high, low, or abnormal based on the range of the test.

### 7.9 Visit Windows

It is expected that all visits should occur according to the protocol schedule. All data will be tabulated per the evaluation visit as recorded on the CRF even if the assessment is outside of the visit window. In data listings, the relative day of all dates will be presented.

### 8 STATISTICAL ANALYSES

### 8.1 Sample Size Determination

Sample size of 104 randomized 1:1 Active to Vehicle based on 80% power to detect 33% IGA response in Active group versus 10% in the Vehicle group, with two-sided test and alpha =0.05. Until mentioned all alpha value is set at 0.05.





### 8.2 Safety Analysis

CLINICAL RESEARCH OPTIMIZED™

Safety analyses will be conducted using the Safety population

### 8.2.1 Primary Safety Endpoint

Assess the safety and tolerability of B244 applied twice daily to the face for 8 weeks in subjects with mild to moderate rosacea.

The reporting of safety data is descriptive and will include all subjects who receive at least one dose of investigational product. The variables for safety endpoints are number of subjects with AEs, SAEs, vital signs measurements, clinical chemistry and hematology. AEs will be summarized based on the frequency of AEs and their severity for all treated subjects. All AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA) and summarized by treatment group. Data will be summarized using preferred term and primary system organ class.

If a subject experiences multiple events that map to a single preferred term, the greatest severity and strongest Investigator assessment of relation to investigational product will be assigned to the preferred term for the appropriate summaries. Should an event have a missing severity or relationship, it will be classified as having the highest severity and/or strongest relationship to investigational product.

Summaries of AEs will include any AEs reported beginning with the first dose of investigational product on Day 1. The occurrence of adverse events will be summarized by treatment group using preferred terms, system organ classifications, and severity. Separate summaries of serious adverse events, adverse events related to investigational product, and events leading to the discontinuation of investigational product will be generated. All adverse events reported will be listed for individual subjects showing both verbatim and preferred terms.

# 8.3 Efficacy Analysis

All efficacy endpoints are exploratory endpoints.

Assessment of Superiority:

- IGA treatment success, defined as "clear" or "almost clear" with a 2-grade improvement in IGA score from baseline to the end of treatment (Week 8).
- CEA treatment success, defined as "clear" or "almost clear" with a 2-grade improvement in CEA score from baseline to the end of treatment (Week 8).

Superiority will be based on the proportion of subjects for whom treatment was successful. The comparison will be through a continuity-corrected Z-tests. The Evaluable Period for the outcome variables will be weeks 1, 4, 8 and 12. The superiority of the drug over the vehicle will be tested at week 8 based on the probability of





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN


> improvement from baseline with a continuity-corrected Z-tests comparing the change from baseline of treatments vs Placebo. For all other evaluable periods, descriptive statistics for the change from baseline will be shown.

> The null and alternative statistical hypotheses for the primary effectiveness endpoints are given by:

> (Ho): The null hypothesis is that the probability of improving (baseline to week 8) with drug T (PrT) is less than or equal to the probability of improving with vehicle (PrV).

```
H o :
       PrT
                -PrPV = VV:
                             PrT
```

(Ha): The alternative hypothesis is that the probability of improving with drug T (PrT) is greater than to the probability of improving with vehicle (PrV).

```
Ha: PrT > PrV; PrT - PrV = 0
```

For testing the superiority, the following SAS code will be used:

```
proc freq data = dataset;
tables treat*outcome/riskdiff (equal);
run;
```

Change of Skindex 16 patient reported outcome from Baseline to Week 1, Week 4, Week 8 and Week 12

The change from baseline score of Skindex-16 will be compared among treatments at Week 12 using an ANOVA, to test the Skindex 16 score change from Baseline to Week 12 for the two treatments. Also, descriptive stats will be used to assess the change from Baseline to Week 1, 4, 8 & 12.

- Change of IGA score at Baseline to Week 1, Week 4, Week 8 and Week 12.
- Change of CEA score at Baseline to Week 1, Week 4, Week 8 and Week 12.
- Change of PSA score at Baseline to Week 1, Week 4, Week 8 and Week 12.

Descriptive stats will be used to show the change from Baseline to Week 1, 4, 8 & 12.

Supplemental Analysis Supplemental analysis will be performed based on any IGA or CEA improvement from Baseline including p-values for the change from Baseline to Week 8 within each treatment group, and IGA and CEA for the subgroup of patients that had a baseline IGA or CEA of 3.

#### 8.4 **Sensitivity Analysis**

A sensitivity analysis will be performed by Multiple Imputation Regression Analysis using the following factors: treatment, age, gender, race, baseline IGA, baseline CEA, baseline





Version 2

02-Apr-19

Protocol: RB244-001 STATISTICAL ANALYSIS PLAN

PSA, smokers/non-smokers and the results of the same variable from previous visits. The Proc MI SAS code will be used to perform the analysis based on the mentioned factors.

### 9 REFERENCES

- Protocol Number: RB244-001, VER 4.0 "A Vehicle-Controlled, Double-Blind, Randomized Phase II Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects with Mild to Moderate Rosacea."
- Wang, Wei. (1988, October 28). Calculating Age in One Line of Code. Paper presented at annual meeting of Northeast SAS Users Group, New York, New York. Paper retrieved from http://www.lexjansen.com/nesug/nesug01/cc/cc4022.pdf.
- DE MARS, A. (2018). "Mixed Reviews": An Introduction to Proc Mixed. Retrieved from <a href="http://www.hawaii.edu/hisug/pdf/AnnMariaprocmixed.pdf">http://www.hawaii.edu/hisug/pdf/AnnMariaprocmixed.pdf</a>
- Moser, E. (2018). Repeated Measures Modeling with PROC MIXED. Retrieved from http://www2.sas.com/proceedings/sugi29/188-29.pdf





# 10 APPENDIX

# 10.1 APPENDIX A: Tables

# **10.1.1 General**

| Display Number | Title | Population | Unique/Repeat |
|---|---|---|---|
| 14.1.1.1 | Subject Enrollment and Disposition | All Subjects | Unique |
| 14.1.1.2 | Subject Enrollment and Disposition | Enrolled Subjects | Unique |
| 14.1.1.3 | Analysis Population and Exclusions | All Subjects | Unique |
| 14.1.2.1 | Summary of Protocol Deviations (PD)/Violations (PV) | mITT | Unique |
| 14.1.2.2 | Summary of Protocol Deviations (PD)/Violations (PV) | Safety | Repeat |
| 14.1.3.1 | Summary of Demographic and Baseline<br>Characteristics | mITT | Unique |
| 14.1.3.2 | Summary of Demographic and Baseline<br>Characteristics | PP | Repeat |
| 14.1.3.3 | Summary of Demographic and Baseline<br>Characteristics | Safety | Repeat |
| 14.1.4.1 | Summary of Vital Sign | mITT | Unique |
| 14.1.4.2 | Summary of Vital Sign | PP | Repeat |
| 14.1.4.3 | Summary of Vital Sign | Safety | Repeat |
| 14.1.5.1 | Summary of Physical Examination | mITT | Unique |
| 14.1.5.2 | Summary of Physical Examination | PP | Repeat |
| 14.1.5.3 | Summary of Physical Examination | Safety | Repeat |
| 14.1.6 | Summary of Study Drug Accountability: Dose Dispensed & Collected by Visit | Safety | Unique |
| 14.1.7.1 | Summary of Study Drug Compliance | Safety | Unique |
| 14.1.7.2 | Summary of Percent Compliance based on<br>Cumulative Net Weight of Study Drug | Safety | Unique |
| 14.1.8 | Summary of Prior or Concomitant<br>Medications | Safety | Unique |
| 14.1.9 | Summary of Medical History | Safety | Unique |
| 14.1.10 | Summary of Substance Abuse | Safety | Unique |
| 14.1.11 | Summary of Dairy Details | Safety | Unique |






### STATISTICAL ANALYSIS PLAN

Version 2 02-Apr-19

Table 14.1.1.1 Subject Enrollment and Disposition

# All Subjects

| | B244 Topical Spray | Placebo | All Patients |
|---|---|---|---|
| Disposition | n (%) | n (%) | n (%) |
| Screened | XX | XX | xx (xx.x) |
| Randomized | xx | XX | xx (xx.x) |
| Treated | xx | XX | xx (xx.x) |
| Completed Study | xx | xx | xx (xx.x) |
| Discontinued | xx | xx | xx (xx.x) |
| Screen Failure | xx | XX | xx (xx.x) |
| Withdrawal of consent | xx | xx | xx (xx.x) |
| In the opinion of the Investigator, it is not in the subject's best interests to continue in the study | xx | XX | xx (xx.x) |
| Pregnancy | XX | XX | xx (xx.x) |
| Occurrence of an Adverse Event (AE) or | XX | xx | xx (xx.x) |
| Serious Adverse Event (SAE), which, in the | | | |
| opinion of the Investigator warrants | | | |
| discontinuation of the subject from the study | | | |
| The subject is lost to follow-up | XX | XX | xx (xx.x) |
| Other | XX | xx | xx (xx.x) |

NOTE: The percentages are based on the

Snapshot Data DD-MMM-YYYY

number of All subjects.
Subjects may have more than one reason for discontinuation, and they are

counted more than once.

Source: <Dataset>

Program Name: <Pgm name>






### STATISTICAL ANALYSIS PLAN

Version 2 02-Apr-19

# Table 14.1.1.2 Subject Enrollment and Disposition

# **Enrolled Subjects**

| Disposition | B244 Topical Spray<br>n (%) | Placebo<br>n (%) | All Patients n (%) |
|---|---|---|---|
| Randomized | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treated | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed Week 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed Week 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed Week 8 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed Week 12 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal of consent | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| In the opinion of the Investigator, it is not in the subject's best interests to continue in the study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Occurrence of an Adverse Event (AE) or Serious Adverse Event (SAE), which, in the opinion of the Investigator warrants discontinuation of the subject from the study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| The subject is lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) |

NOTE: The percentages are based on the number of Randomized subjects.

Subjects may have more than one reason for discontinuation, and they are

counted more than once.

Snapshot Data DD-MMM-YYYY

Source: <Dataset> Program Name: <Pgm name>






### STATISTICAL ANALYSIS PLAN

Version 2 02-Apr-19

# Table 14.1.1.3 Analysis Population and Exclusions All Subjects

| Number of Subjects | B244 Topical Spray n (%) | Placebo<br>n (%) | All Patients n (%) |
|---|---|---|---|
| Enrolled | XX | XX | XX |
| Randomized | xx | XX | XX |
| Included in Safety Population | XX | XX | xx (xx.x%) |
| Reasons for Exclusion from Safety Population | | | |
| | xx | XX | xx (xx.x%) |
| | xx | XX | xx (xx.x%) |
| Included in Full Analysis Set | XX | XX | xx (xx.x%) |
| Reasons for Exclusion from Safety Population | | | |
| | xx | XX | xx (xx.x%) |
| Included in Per Protocol Population | XX | XX | xx (xx.x%) |
| Reasons for Exclusion from Per Protocol Population | | | |
| Lost To Follow Up | XX | XX | xx (xx.x%) |
| Major Deviation | XX | XX | xx (xx.x%) |
| Not 50% Ip Compliant | XX | XX | xx (xx.x%) |
| Screen Failure | XX | XX | xx (xx.x%) |
| Withdrawal of Consent By Subject | xx | XX | xx (xx.x%) |

NOTE: The percentages are based on the number of All subjects.

Snapshot Data DD-MMM-YYYY

Program Name: <Pgm name>

Source: <Dataset>





# Table 14.1.2.1 Summary of Protocol Deviations (PD)/Violations (PV) mITT Population

| | | B244 Topical | | All |
|---|---|---|---|---|
| | Deviation/Violation | Spray | Placebo | Patients |
| Deviation/Violation | Category | n (%) | n (%) | n (%) |
| Description of | "Major" or | n (%) | n (%) | n (%) |
| Violation/deviation | "Minor" | XX | XX | XX |

NOTE: The percentages are based on the number of ITT Population.

Source: <Dataset> Snapshot Data DD-MMM-YYYY

Program Name: <Pgm name>

Repeat for Safety Population

Table 14.1.3.1 Summary of Demographic and Baseline Characteristics mITT Population

| Variable | Statistic | B244 Topical Spray<br>n (%) | Placebo<br>n (%) | All Patients n (%) |
|---|---|---|---|---|
| Age | N | XX | XX | XX |
| _ | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | xx.x(xx.xxx) |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Sex | | | | |
| Male | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Female | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Ethnicity | | | | |
| Hispanic or Latino | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Not Hispanic or Latino | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Race | | | | |
| American Indian or | | | | |
| Alaskan Native | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Asian | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Black or African | | | | |
| American | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Native Hawaiian or | | | | |
| Other Pacific Islander | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |






| | | B244 Topical Spray | Placebo | All Patients |
|----------|-----------|--------------------|-----------|--------------|
| Variable | Statistic | n (%) | n (%) | n (%) |
| White | N (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

NOTE: The percentages are based on the number of ITT Population.

Snapshot Data DD-MMM-YYYY

Program Name: <Pgm name>

Source: <Dataset>

Repeat for PP and Safety population

Table 14.1.4.1 Summary of Vital Signs, mITT Population

| F.7. *. | V. 10. | G | B244 Topical<br>Spray | Placebo | All Patients |
|---|---|---|---|---|---|
| Visit | Vital Sign | Statistic | n (%) | n (%) | n (%) |
| Baseline | Height | N<br>N | XX | XX | XX |
| | | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | XX.X |
| | | | | | (xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Weight | N | XX | XX | XX |
| | | | | | XX.X |
| | | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | (xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Temperature | N | XX | XX | XX |
| | | | | | XX.X |
| | | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | (xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Heart Rate | N | XX | XX | XX |
| | | | | | XX.X |
| | | Mean (SD) | xx.x(xx.xxx) | xx.x (xx.xxx) | (xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Systolic BP | N | XX | XX | XX |
| | • | | | | XX.X |
| | | Mean (SD) | xx.x (xx.xxx) | xx.x (xx.xxx) | (xx.xxx) |






| | | | B244 Topical | | |
|---|---|---|---|---|---|
| | | | Spray | Placebo | All Patients |
| Visit | Vital Sign | Statistic | n (%) | n (%) | n (%) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Diastolic BP | N | XX | XX | XX |
| | | | | | XX.X |
| | | Mean (SD) | xx.x (xx.xxx) | xx.x (xx.xxx) | (xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Repeat for every visit showing | | | | | |
| Change from | | | | | |
| Baseline Baseline | | | | | |
| | | | | | Snapshot Data |

NOTE: The percentages are based on the number of ITT Population.

CRF pages 05-06

DD-MMM-YYYY

Source: <Dataset>

Program Name: <Pgm name>

Repeat for PP and Safety population

Table 14.1.5.1 Summary of Physical Examination, mITT Population

| | | | B244 Topical | | |
|---|---|---|---|---|---|
| | | | Spray | Placebo | All Patients |
| Visit | Physical Examination | Statistic | n (%) | n (%) | n (%) |

Baseline

| General Appearance | | | | |
|----------------------|-------|----------|----------|-----------|
| Normal | N (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Abnormal | N (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Heart Cardiovascular | | | | |
| Normal | N (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |






| Joinnachtan | | | | | 02 / ipi 17 |
|---|---|---|---|---|---|
| | | | B244 Topical | | |
| | | | Spray | Placebo | All Patients |
| Visit | Physical Examination | Statistic | n (%) | n (%) | n (%) |
| | Abnormal | N (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Lungs | | | | |
| | Normal | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Abnormal | N (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Gastrointestinal | , , | , , , | , , | |
| | Normal | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Abnormal | N (%) | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| | Ear/Nose/Throat | , , | , , , | , , | , , |
| | Normal | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Abnormal | N (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Extremities | , , | , , , | , , | , , |
| | Normal | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Abnormal | N (%) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| | Skin | ` , | , , , | . , | ` , |
| | Normal | N (%) | xx(xx.x) | xx (xx.x) | xx(xx.x) |
| | Abnormal | N (%) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Repeat for | | ` , | ` ′ | ` / | • • |
| every week | | | | | |
| | percentages are based on the | ; | | Snapshot Da | ta DD-MMM-YYY |
| 1 | C | | | | |

number of ITT Population.

CRF pages 05-06

Source: <Dataset> Program Name: <Pgm name>

Repeat for PP and Safety populations

Table 14.1.6
Summary of Study Drug Accountability: Dose Dispensed & Collected by Visit
Safety Population
B244 Topical

| | | | Spray | Placebo | All Patients |
|---|---|---|---|---|---|
| Weight of the Dose | Visit | Statistic | n (%) | n (%) | n (%) |
| Dose Dispensed | Baseline | N | XX | XX | XX |
| | | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | xx.x(xx.xxx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Repeat for Dose Collected by Visits





Protocol: RB244-001 STATISTICAL Confidential

STATISTICAL ANALYSIS PLAN

Version 2 02-Apr-19

N: Number of Patients

. . .

CRF pages 28-30

Snapshot Data DD-MMM-YYYY
Program Name: <Pgm name>

Mean(SD): Mean (Standard Deviation),CV: Coefficient of Variance..

Source: <Dataset>

Table 14.1.7.1 Summary of Study Drug Compliance Safety Population

| | | B244 Topical | | All |
|---|---|---|---|---|
| | | Spray | Placebo | Patients |
| | Statistic | n (%) | n (%) | n (%) |
| Number of Subjects wit | :h | | | |
| Compliance | | | | |
| Yes | N (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| No | N (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| If No, Applications<br>Missed | | | | |
| Missed Applications | N | XX | XX | XX |
| | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | XX.X |
| | | | | (xx.xxx) |
| | CV | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, |
| | | | | XX.X |
| Applications: Number of | of applications per pa | atients/day | Snanshot Da | ata DD-MMM- |

Applications: Number of applications per patients/day (expected 4 Pumps twice a Day)

Snapshot Data DD-MMM-YYYY

CRF pages 30

Compliance: The expected amount of study drug used

Program Name: <Pgm

per week is approximately 7.84 g/week for 8 sprays/application per day

Source: <Dataset>

name>

T 11 141 7 0

Table 14.1.7.2 Summary of Percent Compliance based on Cumulative Net Weight of Study Drug Safety Population







| | | B244 Topical | | • |
|---|---|---|---|---|
| | | Spray | Placebo | All Patients |
| | Statistic | n (%) | n (%) | n (%) |
| Cumulative Net Weight | | | | |
| of Study Drug | | | | |
| , 0 | N | XX | XX | XX |
| | Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | xx.x(xx.xxx) |
| | CV | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Percent Compliance | | | | |
| greater than 50% | | | | |
| Yes | N (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| No | N (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Applications: Number of applications per patients/day (expected 4 Pumps twice a Day)

Snapshot Data DD-MMM-YYYY

CRF pages 30

The cumulative amount of study drug exposure will be estimated by calculating the difference between the weight of the 2 bottles of drug at the time the drug was dispensed at Baseline/Week 4 and the weight of the 2 bottles at Week 4/Week 8. Differences will be summed together.

Program Name: <Pgm name>

Source: <Dataset>

Table 14.1.8 Summary of Prior or Concomitat Medications, Safety Population

| WHO-DD ATC Class Level 1 | B244 Topical | | |
|---|---|---|---|
| WHO-DD ATC Class Level 2 | Spray | Placebo | All Patients |
| WHO-DD Preferred Term | n (%) | n (%) | n (%) |
| Number of subjects with at least one prior medication | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| WHO-DD ATC Class Level 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>%</sup> Compliance: The net weight of study drug divided by 1.12g /Day \* Number of Days in the Study







|--------------------------|---------------------------|-----------|-----------|
| WHO-DD ATC Class Level 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| WHO-DD Preferred Term 1 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD Preferred Term 2 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| etc. | | | |
| WILLO DD ATO OL I III | | ( ) | ( ) |
| WHO-DD ATC Class Level 1 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD ATC Class Level 2 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD Preferred Term 1 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| WHO-DD Preferred Term 2 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| etc. | | | |

NOTE: The percentages are based on the

Snapshot Data DD-MMM-YYYY

number of Safety Population.

CRF page 11 Source: <Dataset>

Program Name: <Pgm name>

Table 14.1.9 Summary of Medical History Safety Population

| B244 Topical<br>Spray | Placebo | All Patients |
|---|---|---|
| n (%) | n (%) | n (%) |
| xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx(xx.x) | xx(xx.x) | xx(xx.x) |
| xx (xx.x) | xx (xx.x) | xx(xx.x) |
| xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Spray<br>n (%)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | Spray n (%) Placebo n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) |

NOTE: The percentages are based on the number of Safety Population.

Snapshot Data DD-MMM-YYYY

CRF pages

Source: <Dataset> Program Name: <Pgm name>

Table 14.1.10 Summary of Substance Abuse Safety Population

B244
Topical Placebo All Patients
Statistics Spray N (xxx) N (xxx)





| | | N (xxx) | | |
|---|---|---|---|---|
| Total Number of Substance Abuse | n | xx | XX | XX |
| | | XX | XX | XX |
| | | XX | XX | XX |
| Number of Subjects with Substance<br>Abuse History | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| • | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | xx(xx.x) | xx(xx.x) | xx(xx.x) |

NOTE: The percentages are based on the number of Safety Population.

Snapshot Data DD-MMM-YYYY

CRF pages

Source: <Dataset> Program Name: <Pgm name>

Table 14.1.11 Summary of Diary Details Safety Population

| | Statistics | B244 Topical<br>Spray<br>N (xxx) | Placebo<br>N (xxx) | All Patients<br>N (xxx) |
|---|---|---|---|---|
| Number of Subjects with diary Dispensed<br>Number of Subjects with diary Collected | n<br>n | XX<br>XX<br>XX | XX<br>XX<br>XX | XX<br>XX<br>XX |
| Number of Subjects with Sunscreen use<br>Number of Subjects with Makeup use | n (%)<br>n (%) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |

NOTE: The percentages are based on the number of Safety Population.

Snapshot Data DD-MMM-YYYY

CRF pages

Source: <Dataset> Program Name: <Pgm name>





# 10.1.2 Efficacy

| Display Number | Title | Population | Unique/Repeat |
|---|---|---|---|
| 14.2.1.1 | Change from baseline in IGA score by Visit | mITT | Unique |
| 14.2.1.2 | Change from baseline in IGA score by Visit | PP | Repeat |
| 14.2.2.1 | Change from baseline in CEA score by Visit | mITT | Repeat |
| 14.2.2.2 | Change from baseline in CEA score by Visit | PP | Repeat |
| 14.2.3.1 | Change from baseline in PSA score by Visit | mITT | Repeat |
| 14.2.3.2 | Change from baseline in PSA score by Visit | PP | Repeat |
| 14.2.4.1 | Summary of Change from baseline in Skindex 16 score by Visit | mITT | Unique |
| 14.2.4.2 | Summary of Change from baseline in Skindex 16 score by Visit | PP | Repeat |
| 14.2.5.1 | Change from baseline in Telangiectasia score by Visit | mITT | Repeat |
| 14.2.5.2 | Change from baseline in Telangiectasia score by Visit | PP | Repeat |
| 14.2.6.1 | Summary of 2-grade improvement in IGA score from baseline to the end of treatment. | mITT | Unique |
| 14.2.6.2 | Summary of 2-grade improvement in IGA score from baseline to the end of treatment | PP | Repeat |
| 14.2.7.1 | Summary of 2-grade improvement in CEA score from baseline to the end of treatment | mITT | Repeat |
| 14.2.7.2 | Summary of 2-grade improvement in CEA score from baseline to the end of treatment. | PP | Repeat |
| 14.2.8.1 | Summary of IGA score of 0/1 at End of Treatment. | mITT | Unique |
| 14.2.8.2 | Summary of IGA score of 0/1 at End of Treatment. | PP | Repeat |
| 14.2.9.1 | Summary of CEA score of 0/1 at End of Treatment. | mITT | Repeat |
| 14.2.9.2 | Summary of CEA score of 0/1 at End of Treatment. | PP | Repeat |
| 14.2.10.1 | Summary of Sensitivity Analysis for<br>Change from Baseline Score of IGA | mITT | Unique |
| 14.2.10.2 | Summary of Sensitivity Analysis for<br>Change from Baseline Score of CEA | mITT | Repeat |
| 14.2.10.3 | Summary of Sensitivity Analysis for<br>Change from Baseline Score of PSA | mITT | Repeat |





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN


# Table 14.2.1.1 Change from baseline in IGA Score by Visit. mITT Population

| | Spray | Placebo | All Patients |
|---------------------------|---------|---------|--------------|
| Visit | N (xxx) | N (xxx) | N (xxx) |
| Week 1 | | | |
| Change from Baseline | | | |
| 1-grade | n (%) | | |
| 2-grade | n (%) | | |
| 3-grade | n (%) | | |
| Repeat for all the visits | | | |

CRF pages Source: <Dataset> Snapshot Data DD-MMM-YYYY

Program Name: <Pgm name>

Repeat for CEA and PSA & Telangiectasia Score for mITT & PP population.

Table 14.2.4.1 Summary of Change from baseline in Skindex 16 score by Visit mITT Population

| | B244 Topical | | |
|---|---|---|---|
| | Spray | Placebo | All Patients |
| Visit | N (xxx) | N (xxx) | N (xxx) |
| Baseline | | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x(xx.xxx) | xx.x (xx.xxx) | xx.x (xx.xxx) |
| CV | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Change from Baseline at Week 1 | | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x(xx.xxx) | xx.x(xx.xxx) | xx.x(xx.xxx) |
| CV | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |






Final Analysis for Week 12

Differences of LS Means x.xxxx SE x.xxxx

CI P-value (x.xxxx, x.xxxx)

SE: Standard Error of the LS Means

CRF pages Source: <Dataset> Snapshot Data DD-MMM-YYYY

Program Name: <Pgm name>

Repeat for PP population.

# Table 14.2.10.1 Summary of Sensitivity Analysis for Change from Baseline Score of IGA mITT Population

| | B244 Topical<br>Spray | Placebo | All Patients |
|---|---|---|---|
| Imputation | N (xxx) | N (xxx) | N (xxx) |
| Imputation#1 | | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x(xx.xxx) | xx.x (xx.xxx) | xx.x (xx.xxx) |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Imputation#2 | | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x(xx.xxx) | xx.x (xx.xxx) | xx.x (xx.xxx) |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Repeat for all imputations | | | |
| Analysis Summary | | | |
| Mean (SD) | | | x.xx, x.xx |
| CI | | | X.XXX |
| P-Value | | | |

SD: Standard Error of the Parameters

CI: Confidence Interval





Repeat for CEA & PSA.

CRF pages
Source: <Dataset>

Snapshot Data DD-MMM-YYYY
Program Name: <Pgm name>

Table 14.2.6.1 Summary of 2-grade improvement in IGA score from baseline to the end of treatment. mITT Population

| | B244 Topical<br>Spray<br>N (xxx) | Placebo<br>N (xxx) | All Patients<br>N (xxx) |
|---|---|---|---|
| Subjects with 2-Grade improvement from Baseline to End of Treatment | n (%) | n (%) | n (%) |
| Risk Difference<br>CI<br>P-value | | | x.xxx<br>(x.xx, x.xx)<br>x.xxxx |

CI: Confidence Interval

Snapshot Data DD-MMM-YYYY

Source: <Dataset>

Program Name: <Pgm name>

Repeat for PP Population and for CEA (mITT & PP).

# Table 14.2.8.1 Summary of IGA score of 0/1 at End of Treatment. mITT Population

| | B244 Topical | | |
|---|---|---|---|
| | Spray | Placebo | All Patients |
| | N(xxx) | N(xxx) | N (xxx) |
| Subjects with Score of 0/1 at End of Treatment | n (%) | n (%) | n (%) |
| Risk Difference<br>CI<br>P-value | | | x.xxx<br>(x.xx, x.xx)<br>x.xxxx |





Protocol: RB244-001 STATISTICAL ANALYSIS PLAN Confidential

Version 2 02-Apr-19

CI: Confidence Interval

Snapshot Data DD-MMM-YYYY

Program Name: <Pgm name>

Source: <Dataset> Repeat for PP Population and for CEA (mITT & PP)

# **10.1.3** Safety

| Display Number | Title | Population | Unique/Repeat |
|---|---|---|---|
| 14.3.1 | Overall Summary of Treatment Emergent<br>Adverse Events | Safety | Unique |
| 14.3.1.1 | Summary of Treatment Emergent Adverse<br>Events by System Organ Class and<br>Preferred Term | Safety | Unique |
| 14.3.1.2 | Summary of Treatment Emergent Adverse<br>Events by System Organ Class, Preferred<br>Term and Severity | Safety | Repeat |
| 14.3.1.3 | Summary of Treatment Emergent Adverse<br>Events by System Organ Class, Preferred<br>Term and Relationship to Study Drug | Safety | Repeat |
| 14.3.2 | Summary of Serious Adverse Events by<br>System Organ Class and Preferred Term | Safety | Repeat |
| 14.3.3 | Summary of Deaths | Safety | Unique |

Table 14.3.1 Overall Summary of Treatment Emergent Adverse Events. Safety Population

| | | B244 Topical | | |
|---|---|---|---|---|
| | g | Spray | Placebo | All Patients |
| | Statistics | n (%) | n (%) | n (%) |
| Total Number of TEAEs | N | XX | XX | xx |
| Total Number of TESAEs | N | XX | XX | XX |
| Number of Subjects with: | | | | |
| At Least One TEAE | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| At Least One Related TEAE | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| At Least One Severe (Grade 3) TEAE | n (%) | xx (xx.x) | xx(xx.x) | xx(xx.x) |
| At Least One TEAE Leading to Discontinuation | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| At Least One TEAE Leading to Death | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| At Least One TESAE | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| At Least One Related TESAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |





NOTE: The percentages are based on the

Snapshot Data DD-MMM-YYYY

number of Safety Population.

CRF pages

Source: <Dataset> Program Name: <Pgm name>

Table 14.3.1.1
Overall Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred
Term
Safety Population

| | Statistics | B244 Topical<br>Spray<br>n (%) | Placebo<br>n (%) | All Patients<br>n (%) |
|---|---|---|---|---|
| Total Number of TEAEs | n | XX | xx | XX |
| Number of Subjects with at Least One TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #1 Preferred Term #1 Preferred Term #2 Preferred Term #3 etc. | n (%)<br>n (%)<br>n (%)<br>n (%) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| System Organ Class #2 Preferred Term #1 Preferred Term #2 Preferred Term #3 etc. | n (%)<br>n (%)<br>n (%)<br>n (%) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

NOTE: The percentages are based on the

Snapshot Data DD-MMM-YYYY

number of Safety Population.

CRF pages

Source: <Dataset>

Program Name: <Pgm name>

Table 14.3.1.2

Overall Summary of Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Severity

Safety Population

| | Statistics | Severity | B244 Topical<br>Spray<br>N (xxx) | Placebo<br>N (xxx) | All Patients<br>N (xxx) |
|---|---|---|---|---|---|
| Total Number of TEAEs | n | Mild<br>Moderate | xx<br>xx | XX<br>XX | xx<br>xx |







| Protocol: RB244-001<br>Confidential | STATISTICAL ANALYSIS PLAN | | | | Version 2<br>02-Apr-19 |
|---|---|---|---|---|---|
| | | Severe | XX | XX | XX |
| | | Total | xx | XX | XX |
| Number of Subjects with at Least One TEAE | n (%) | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Moderate | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| | | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #1 | n (%) | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| , | . , | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #1 | n (%) | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | . , | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Total | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| etc. | | | , | | , |
| NOTE: The percentages are based on the number of Safety Population. Subject has more than 1 AE on a Preferred term, then, it is counted only once on the | | F pages | Snapshot Data I<br>Program Na | DD-MMM-YY<br>ame: <pgm na<="" td=""><td></td></pgm> | |
| highest severity. | | arce: | | | |

Table 14.3.1.3

Overall Summary of Treatment Emergent Adverse Events by System Organ Class, Preferred
Term, and Relationship to Study Drug
Safety Population

| | Statistics | Relationship | B244<br>Topical<br>Spray<br>N (xxx) | Placebo<br>N (xxx) | All Patients N (xxx) |
|---|---|---|---|---|---|
| Total Number of TEAEs | n | Not Related<br>Related<br>Total | xx<br>xx<br>xx | xx<br>xx<br>xx | xx<br>xx<br>xx |
| Number of Subjects with at Least One TEAE | n (%) | Not Related<br>Related<br>Total | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | ) xx (xx.x) |





| Protocol: RB244-001 | STATIST | TATISTICAL ANALYSIS PLAN | | | ersion 2 |
|---|---|---|---|---|---|
| Confidential | | | | 02- | -Apr-19 |
| System Organ Class #1 | n (%) | Not Related | d xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Related | xx(xx.x) | xx (xx.x) | xx(xx.x) |
| | | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #1 | n (%) | Not Related | d xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Related | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | | Total | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| etc. | | | | | |
| | CF | RF pages | Snapshot Data DD-N | MMM-YYYY | |
| NOTE: The percentages are based on the | So | ource: | Program Name: | <pgm name=""></pgm> | |
| number of Safety Population. | <[ | Dataset> | - | - | |

Table 14.3.2 Summary of Serious Adverse Events by System Organ Class and Preferred Term Safety Population

| | | | B244 Topical<br>Spray | Placebo | All<br>Patients |
|---|---|---|---|---|---|
| | Statistics | Relationship | N (xxx) | N (xxx) | N (xxx) |
| Total Number of SAEs | n | Yes | XX | XX | XX |
| Total Trainion of STIES | | No | XX | XX | XX |
| | | Total | XX | XX | XX |
| Number of Subjects with at<br>Least One SAE | n (%) | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | No | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| | | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #1 | n (%) | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | No | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Duefermed Town #1 | ·· (0/) | Vas | () | () | () |
| Preferred Term #1 | n (%) | Yes | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| | | No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Total | xx (xx.x) | xx(xx.x) | xx(xx.x) |
| etc. | | | | | |
| | CRF pages | 3 | Snapshot Data DD-l | MMM-YYYY | |





Program Name: <Pgm name>


NOTE: The percentages are based

on the number of Safety

Population. Source: <Dataset>

Table 14.3.3 Summary of Deaths Safety Population

B244 Topical Spray Placebo All Patients Statistics N(xxx)N(xxx)N(xxx)Number of deaths xx (xx.x%) xx (xx.x%) n (%) xx(xx.x%)Related to disease under study n (%) xx(xx.x%)xx(xx.x%)xx(xx.x%)

AE outcome = death n (%) xx (xx.x%) xx (xx.x%) xx (xx.x%) Related to disease under study n (%) xx (xx.x%) xx (xx.x%) xx (xx.x%) and AE outcome = death

CRF pages Snapshot Data DD-MMM-YYYY

Program Name: <Pgm name>

NOTE: The percentages are based on the number of Safety Population.

Source: <Dataset>

# 10.2 APPENDIX B: Listings

| Display Number | Title | Population |
|---|---|---|
| Listing 16.2.1.1 | Subject Enrollment and Disposition by Study Site | All Subjects |
| Listing 16.2.1.2 | Protocol Deviations (PD)/Violations (PV) | Randomized |
| Listing 16.2.1.3 | Demographic Characteristics | Randomized |
| Listing 16.2.1.4 | Vitals Signs by Subject and Visit | Safety |
| Listing 16.2.1.5 | Physical Examination by Subject | Safety |
| Listing 16.2.1.6 | Drug Exposure and Compliance | Safety |
| Listing 16.2.1.8 | Prior and Concomitant Medications | Safety |
| Listing 16.2.1.9 | Medical History | Safety |
| Listing 16.2.2.1 | IGA score by Subjects and Visits | Randomized |
| Listing 16.2.2.2 | CEA score by Subjects and Visits | Randomized |
| Listing 16.2.2.3 | PSA score by Subjects and Visits | Randomized |
| Listing 16.2.2.4 | Skindex-16 score by Subjects and Visits | Randomized |
| Listing 16.2.2.5 | Telangiectasia Evaluation by Subjects and Visits | Randomized |
| Listing 16.2.2.6 | Fitzpatrick Classification by Subjects and Visits | Randomized |
| Listing 16.2.3.1 | Treatment Emergent Adverse Events by System Organ | Safety |
| | Class, Preferred Term, Severity and Relationship to | |
| | Study Drug | |






| Communication | 0 <b>2</b> 1101 17 | |
|---|---|---|
| Listing 16.2.3.2 | Serious Adverse Events by System Organ Class and Preferred Term | Safety |
| Listing 16.2.3.3 | Deaths | Safety |
| Listing 16.2.4.1 | Hematology Parameters | Safety |
| Listing 16.2.4.2 | Clinical Chemistry Parameters | Safety |
| Listing 16.2.4.3 | Urinalysis Parameters | Safety |

# 10.3 APPENDIX C: Figures

| Display Number | Title | Population |
|---|---|---|
| Figure 14.2.1.1 | Frequency table Change from baseline for IGA score by Visit | mITT |
| Figure 14.2.1.2 | Frequency table Change from baseline for IGA score by Visit | PP |
| Figure 14.2.2.1 | Frequency table Change from baseline for CEA score by Visit | mITT |
| Figure 14.2.2.2 | Frequency table Change from baseline for CEA score by Visit | PP |
| Figure 14.2.3.1 | Frequency table Change from baseline for PSA score by Visit | mITT |
| Figure 14.2.3.2 | Frequency table Change from baseline for PSA score by Visit | PP |
| Figure 14.2.4.1 | Box Plot of Skindex16 score by Visit | mITT |
| Figure 14.2.4.2 | Box Plot of Skindex16 score by Visit | PP |
| Figure 14.2.8.1 | Bar Plot of IGA & CEA score at End of Treatment | mITT |
| Figure 14.2.8.2 | Bar Plot of IGA & CEA score at End of Treatment | PP |
| Figure 14.2.9.1 | Bar Plot of IGA & CEA score for more than 2-grade improvement from Baseline to End of Treatment. | mITT |
| Figure 14.2.9.2 | Bar Plot of IGA & CEA score for more than 2-grade improvement from Baseline to End of Treatment. | PP |